# STATISTICAL ANALYSIS PLAN

Study Title: Safety, Tolerability, Efficacy and Dose Response of GLS-

1027 in the Prevention of Severe Pneumonitis caused by

SARS-CoV-2 Infection

Name of Test Drug: GLS-1027

**Study Number:** GLS27-005

**Protocol Version:** 5.0

**Protocol Date:** 11 Aug 2021

**Analysis Plan Version:** 1.0

**Analysis Plan Date:** 03 Dec 2021

Analysis Plan Author: Catalyst Clinical Research, LLC

CONFIDENTIAL AND PROPRIETARY INFORMATION

# SIGNATURE PAGE

Signature

Date 3 December 2021

Dr. Joel Maslow

Chief Medical Officer

GeneOne Life Science Inc.

-DocuSigned by:

Susan E. Spruill

U

Signer Name: Susan E. Spruill Signing Reason: I approve this document Signing Time: 05-Dec-2021 | 7:53:56 AM CST -6B44CB45B7954FD5B700ED25E98AB084

sec 11c

05-Dec-2021

Signature

Date

Susan E. Spruill, MS, PStat®

Statistical Consultant

Applied Statistics and Consulting

-DocuSigned by:

Ahmed Tarig



Signer Name: Ahmed Tariq Signing Reason: I am the author of this document Signing Time: 03-Dec-2021 | 3:23:04 PM EST

-8A9AFFC7511B48049134C7E9728C3D84

03-Dec-2021

Signature

Date

Ahmed Tariq, MS

Biostatistician

Catalyst Clinical Research, LLC

| LIS | T OF A | ABBREVIATIONS | 4 |
|-----|--------|-------------------------------------------------------|----|
| 1. | INTR | RODUCTION | 5 |
| 2. | STUI | DY OBJECTIVES | 5 |
| | 2.1. | Primary Objectives | 5 |
| | 2.2. | Exploratory Objectives | 5 |
| 3. | STUI | DY DESIGN AND PLAN | 6 |
| 4. | DETE | ERMINATION OF SAMPLE SIZE | 8 |
| 5. | GENI | ERAL ANALYSIS CONSIDERATIONS | 8 |
| 6. | ANA | LYSIS POPULATIONS | 9 |
| | 6.1. | Intent-to-treat (ITT) Population | 9 |
| | 6.2. | Modified Intent-to-treat (mITT) Population | |
| | 6.3. | Safety Population | |
| | 6.4. | Per-protocol (PP) Population | |
| 7. | STUI | DY POPULATION | 9 |
| | 7.1. | Subject Disposition | 9 |
| | 7.1. | Protocol Deviations | |
| | 7.3. | Demographics and Baseline Characteristics | |
| | 7.4. | Medical History | |
| | 7.5. | Prior and Concomitant Medications | |
| | 7.6. | Study Drug Exposure | |
| | 7.7. | Blood Collection for Pharmacokinetic and PBMC Results | |
| 8. | EFFI | CACY ANALYSES | 11 |
| | 8.1. | Definition of the Primary Efficacy Endpoint | 11 |
| | 8.2. | Analysis of the Primary Efficacy Endpoint | |
| | 8.3. | Definition of the Exploratory Efficacy Endpoints | |
| | 8.4. | Analysis of the Exploratory Efficacy Endpoints | |
| 9. | SAFF | ETY ANALYSES | 13 |
| | 9.1. | Adverse Events | 13 |
| | | 9.1.1. Severity | |
| | | 9.1.2. Relationship | 13 |
| | | 9.1.3. Serious Adverse Events | 13 |
| | | 9.1.4. Treatment-Emergent Adverse Events (TEAEs) | |
| | | 9.1.4.1. Definition of Treatment-Emergent | |
| | | 9.1.4.2. Incomplete Dates | |
| | 0.5 | 9.1.5. Summaries of Adverse Events | |
| | 9.2. | Clinical Laboratory Evaluations | |
| | 9.3. | Vital Signs | |
| | 9.4. | ECG Results | |
| | 9.5. | Physical Exam | |
| | 9.6. | Urine Pregnancy Test | 16 |

| APPENDIX A: PRESENTATION OF DATA AND PROGRAMMING SPECIFICATIONS | 17 |
|-------------------------------------------------------------------|----|
| APPENDIX B: TABLE OF CONTENTS FOR STATISTICAL TABLES AND LISTINGS | 20 |
| APPENDIX C: TABLE LAYOUTS | 26 |
| APPENDIX D: FIGURE LAYOUTS | 63 |
| APPENDIX E: LISTING LAYOUTS | 66 |

### LIST OF ABBREVIATIONS

AE adverse event

ATC Anatomical Therapeutic Chemical

BMI body mass index
bpm beats per minute
CRF case report form
CSR Clinical Study Report
DBP diastolic blood pressure
ECG electrocardiogram
ET early termination

FDA Food and Drug Administration

GI gastrointestinal

HBsAg hepatitis B surface antigen

HCV hepatitis C virus

ICH International Conference on Harmonisation

IP Investigational Product

ITT Intent-to-Treat

MedDRA Medical Dictionary for Regulatory Activities

OTC over-the-counter

PEEP Positive End-Expiratory Pressure

PT preferred term

SAE serious adverse event
SBP systolic blood pressure
SD standard deviation
SOC system organ class

TLFs tables, listings, and figures ULN upper limit of normal WHO World Health Organization

#### 1. INTRODUCTION

This document outlines the statistical methods to be implemented during the analyses of data collected within the scope of GeneOne Life Science Inc.'s Protocol GLS27-005 [Safety, Tolerability, Efficacy and Dose Response of GLS-1027 in the Prevention of Severe Pneumonitis caused by SARS-CoV-2 Infection]. The purpose of this plan is to provide specific guidelines from which the statistical analyses will proceed. Any deviations from this plan will be documented in the clinical study report (CSR).

The reader is referred to the following complementary documents:

- Protocol GLS27-005, version 5.0, dated 11 Aug 2021
- Case Report Form (CRF), version 1.05, dated 08 Feb 2021
- Data Management Plan, version 1.0, dated 04 Feb 2021

#### 2. STUDY OBJECTIVES

# 2.1. Primary Objectives

The primary objectives of the study are to evaluate the following:

- Incidence of serious adverse events relative to treatment group
- Incidence of treatment failure within 28 days from enrollment

# 2.2. Exploratory Objectives

The exploratory objectives are:

- Assess the number of days requiring ICU care relative to treatment group.
- Assess the number of days of NIV, high-flow O2 or mechanical ventilation relative to treatment group.
- Assess incidence of WHO COVID-19 Classification levels relative to baseline serum IL-6 level.
- Assess incidence of WHO COVID-19 Classification levels relative to baseline serum ferritin level.
- Assess incidence of WHO COVID-19 Classification levels relative to baseline CRP
- Assess trough level of GLS-1027 relative to serum creatinine.
- Assess the maximal level of Positive End-Expiratory Pressure (PEEP) for subjects who are intubated relative to treatment group.
- Assess the number of days of PEEP > 5 cm H2O for subjects who are intubated relative to treatment group.
- Assess change in WHO COVID-19 Classification level at Day 28 from enrollment, relative to group.
- Assess SARS-CoV-2 IgM antibody responses relative to treatment group.

#### 3. STUDY DESIGN AND PLAN

This is a Phase II, randomized, double-blind, placebo-controlled study to assess 2 dose levels of GLS-1027 for the prevention of treatment failure among participants admitted to the hospital with PCR confirmed infection with SARS-CoV-2 (WHO classification 3 or 4). Subjects can be enrolled up to 72 hours from the time of hospital admission.

Participants will be randomized to placebo or GLS-1027 at either 120 mg or 360 mg daily in a 1:1:1 ratio as adjunctive to standard of care based on the hospital COVID-19 treatment algorithm and/or local COVID-19 treatment practices. Participants will be administered study drug for a maximum treatment period of 14 days or until discharge or death, whichever comes first. Primary outcome will be assessment at day 28, with follow-up to continue to Day 56 to document AEs and outcome as to discharge, death, or WHO COVID-19 classification level if subject remains hospitalized.

All subjects will be considered to have completed the study except for the following circumstances:

- Withdrawal of consent from study
- Loss to follow-up
- Stopped study treatment for any reason other than discharge, pregnancy, or decreased renal function

**Table 1: Schedule of Assessments** 

| Tests and Observations | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 28 | 56 <sup>m</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Clinical Evaluations | | | | | | | | | | | | | | | | | |
| Obtain written Informed Consent | Х | | | | | | | | | | | | | | | | |
| Confirm Eligibility Criteria | Х | | | | | | | | | | | | | | | | |
| Demographics | Х | | | | | | | | | | | | | | | | |
| Medical History | Х | | | | | | | | | | | | | | | | |
| Concomitant Medications | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Review Medical Record | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| WHO COVID-19 Classification (Appendix B) | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Safety Evaluations | | | | | | | | | | | | | | | | | |
| Record Adverse Events | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Record AM Vital Signs a | Х | Х | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | |
| Record Hematology <sup>b</sup> | Х | Х | Х | | | Х | | | Х | | | Х | | | Х | | |
| Record Basic Metabolic Panel <sup>c</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | |
| Record liver function studies (LFTs) ° | Х | | | | | Х | | | Х | | | Х | | | Х | | |
| Record other labs <sup>d</sup> (for days available) | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | |
| Record Procalcitonin (baseline value) e | Х | | | | | | | | | | | | | | | | |
| Record admission CXR | Х | | | | | | | | | | | | | | | | |
| Record if care given in ICU setting | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | |
| Record whether nasal O <sub>2</sub> prescribed and dose<br>level (L/min) <sup>f</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | |
| Record whether CPAP prescribed and<br>expiratory pressure <sup>9</sup> | X | X | X | X | X | X | X | Х | Х | X | Х | X | X | Х | X | | |
| Record if mechanically ventilated and level of<br>PEEP, % FiO <sub>2</sub> h | X | X | Х | X | X | X | Х | X | Х | X | Х | X | Х | X | X | | |
| Record if treated by ECMO | X | Х | X | X | X | X | X | X | X | X | X | X | Х | X | Х | | |
| Record admission ECG | Х | | | | | | | | | | | | | | | | |
| Study Related Procedures | | | | | | | | | | | | | | | | | |
| Administer assigned study drug <sup>1</sup> | Х | Х | X | Х | X | Х | Х | Х | X | Х | Х | X | X | Х | | | |
| Perform urine pregnancy test | Х | | | | | | | | | | | | | | | | |
| Perform ECG (12-lead) J | | Х | | | | | Х | | | | | | | | | | |
| Collect serum for CPK, GGT k | Х | | | | | | Х | | | | | | | | | | |
| Collect blood for plasma for PK assessment <sup>1</sup> | | Х | | | | | | | | | | | | | | | |
| Collect blood for plasma for trough drug<br>measurement (AM blood draw) | | Х | Х | Х | | | Х | | | | | | | | | | |
| Collect blood for serum (10mL red top,3 tubes) | Х | | | | | | Х | | | | | | | Х | | | |
| Collect blood for PBMCs (10mL ACD; 3 tubes) <sup>n</sup> | Х | | | | | | Х | | | | | | | Х | | | |
| Blood volume for serum, PBMCs | 60 | | | | | | 70 | | | | | | | 60 | | | _ |

<sup>&</sup>lt;sup>a</sup> Vital signs to be recorded daily to include: temperature, respiratory rate, heart rate, systolic and diastolic blood pressure


<sup>&</sup>lt;sup>b</sup> Hematology labs to be recorded (as collected as part of clinical care) and recorded: Hemoglobin, hematocrit, platelets, neutrophils, band forms, lymphocytes, eosinophils

<sup>&</sup>lt;sup>c</sup> Basic metabolic panel labs: Sodium, potassium, creatinine, BUN, glucose, liver function tests; LFTs include AST, ALT, bilirubin (direct), alkaline phosphatase, LDH, albumin.

<sup>&</sup>lt;sup>d</sup> Other labs to be recorded if performed: Ferritin, CRP, IL-6, troponin, D-dimer

<sup>&</sup>lt;sup>e</sup> Procalcitonin: record only initial measurement or within 48 hours of admission and/or SARS-CoV-2 diagnosis (may be performed prior to date of enrollment)

f Record maximal daily level of O2 by nasal cannula prescribed, if participant is receiving O2 by nasal cannula

<sup>&</sup>lt;sup>g</sup> Record maximal daily level of end expiratory pressure delivered by CPAP prescribed, if participant is receiving CPAP

- <sup>j</sup> Perform a 12-lead ECG on the 2nd day of treatment with study drug between 75 and 90 minutes post-administration on day 2; and on day 15 (± 2 days)
- <sup>k</sup> Serum is collected for CPK and GGT on day 1 and day 7, and weekly thereafter, if values on day 7 are abnormal until return to normal
- <sup>1</sup> PK assessment will be performed for the initial 15 subjects enrolled. Blood (5 ml) will be collected for plasma collection at baseline (pre-treatment), and then at 1, 2, 4, and 8 hr. Trough measurements will be obtained as indicated for all study participants
- <sup>m</sup> The clinical record should be reviewed at Day 28 and Day 56 as relevant to denote date of discharge, date of death, or clinical status (WHO COVID-19 Classification Level); if discharged, subjects should be contacted by telephone to ascertain clinical status.
- <sup>n</sup> PBMCs will be collected at specified sites only

### 4. DETERMINATION OF SAMPLE SIZE

Based on the initial data obtained to date and data in the literature, it is anticipated that approximately 50% of subjects hospitalized with PCR-positive SARS-CoV-2 infections (WHO COVID-19 Classification level 3 or 4) will experience treatment failure at day 28 from enrollment. Treatment failure is defined as progression to WHO COVID-19 classification level of 6 or greater as defined by one or more of the following: the need for high-flow oxygen or non-invasive ventilation, the need for intubation or mechanical ventilation (level 6), the need for ECMO (level 7), or any cause death (level 8); the initiation of a non-study immune modulator; withdrawing consent from the study; becoming lost to follow-up; or discontinuation of treatment for any reason other than renal function or pregnancy. The sample size estimate for this proof of concept is based on Fisher's Exact two-sided test for 2 proportions using NQuery 8 (www.statsols.com). Estimates of admitted patients requiring salvage therapy is unknown, however, the clinical data set who require intubation is a likely subset of those whose condition worsens but do not progress to respiratory compromise.

Although the interim analysis will utilize masked treatment assignments, the O'Brien Fleming group sequential sample size estimation confirms that a single interim look would retain a cumulative exit probability of 70% with a cumulative alpha =0.05 after the final analysis using the target enrollment of 132 (44 per group) to detect a reduction of those reaching the endpoint of treatment failure. This study is not powered to assess statistically significant differences between GLS-1027 doses. A gate-keeping method will be used to compare the highest dose to placebo first and then compare the lower dose if the higher dose shows significant benefit.

### 5. GENERAL ANALYSIS CONSIDERATIONS

The statistical analysis results will be reported using tables, listings, and figures (TLFs). Summaries of continuous variables will display means, standard deviations (SDs), medians, minimums, maximums, and the number of observations. Summaries of categorical variables will display frequency counts and percentages.


<sup>&</sup>lt;sup>h</sup> Record maximal daily level of PEEP and delivered FiO2 by mechanical ventilation, if participant is receiving mechanical ventilation

<sup>&</sup>lt;sup>i</sup> Study drug administration will commence on the day of enrollment if treatment can be administered before 10 pm and then with AM medications thereafter, If, study drug cannot be administered prior to 10 pm on the day of enrollment, then the 1st day of treatment will occur on the day after enrollment.

All analyses will be performed using SAS® Version 9.4 or higher.

A masked interim analysis will be performed when 22 subjects in each group have been assessed for the primary endpoint of treatment failure. The primary goals of this analysis are to review blinded safety to ensure that GLS-1027 has no concerns or causes worsening conditions. Unless safety is of concern, the study will not be stopped for futility and enrollment will continue to the targeted sample size of 132.

### 6. ANALYSIS POPULATIONS

# 6.1. Intent-to-treat (ITT) Population

The ITT Population will include all subjects randomized to a treatment allocation. The ITT population will be used for the summary of all demographic and baseline characteristics and for analysis of the primary outcome of treatment failure. Subjects will be grouped in analyses and summaries based on their randomization allocation.

# 6.2. Modified Intent-to-treat (mITT) Population

The modified intention to treatment (mITT) population includes all participants who are randomized to a treatment allocation, and who have received at least one dose of study drug. The mITT population will be used for the summary and analysis of the primary outcome of treatment failure. Participants will be grouped based on the treatment allocation.

# 6.3. Safety Population

The Safety Population will include all participants in the mITT population. Subjects will be grouped in analyses and summaries based on their actual treatment.

# 6.4. Per-protocol (PP) Population

The PP Population includes all safety subjects who complete the trial by meeting the endpoint of treatment failure or being discharged within 14 days without meeting the endpoint. Subjects will be grouped in analyses and summaries based on their actual treatment. This set will be used as a sensitivity analysis to summarize the primary and other efficacy outcomes.

#### 7. STUDY POPULATION

# 7.1. Subject Disposition

The number and percentage of subjects who were screened and failed screening, who were in each analysis population, who completed the study and who discontinued prior to study completion will be presented by treatment group (GLS-1027 120 mg, GLS-1027 360 mg, and placebo) and overall. Subjects who discontinued prior to completing the study will also be summarized by reason for discontinuation.

Subject disposition will also be listed.


#### 7.2. Protocol Deviations

Protocol deviations with significance will be listed.

# 7.3. Demographics and Baseline Characteristics

Demographics and baseline data, vital signs, medical history, prior and concomitant medications, and treatments will be summarized by means of descriptive statistics: continuous variables as mean, median, SD, minimum/maximum ranges and categorical variables as frequencies and percentages, grouped by treatment arms and overall, based on ITT population. Demographic and baseline characteristics will also be listed.

# 7.4. Medical History

Medical history verbatim terms collected from the CRF will be mapped to system organ classes (SOCs) and preferred terms (PTs) using the Medical Dictionary for Regulatory Activities (MedDRA) (version 23.0).

Summaries (number and percentage of subjects) of medical history by SOC and PT will be provided by treatment and overall.

A listing of medical history will also be provided.

#### 7.5. Prior and Concomitant Medications

A prior medication is defined as a medication that was administered up to 4 months prior to time of enrollment. All other medications will be considered concomitant.

Medication verbatim names collected from the CRF will be mapped to Anatomical Therapeutic Chemical (ATC) Classes and Preferred Names using the World Health Organization's WHODrug Global March 2020 version. Preferred Names will consist of only the base compounds and not the salts (e.g., Naproxen Sodium will be listed only as Naproxen). Concomitant medications will be summarized for each treatment by ATC class and preferred name. Prior and concomitant medications will be listed.

# 7.6. Study Drug Exposure

Exposure summaries of duration of exposure, total number of doses taken, and total number of doses missed will be provided by treatment. Duration of exposure is defined as the date of last dose minus the date of first dose + 1, regardless of if any doses were missed in between. Exposure data will be listed.

### 7.7. Blood Collection for Pharmacokinetic and PBMC Results

Blood collection information (date/time and volume of blood) for PK assessments, trough drug measurements, serum, and PBMCs will be listed.


#### 8. EFFICACY ANALYSES

# 8.1. Definition of the Primary Efficacy Endpoint

The primary endpoint is treatment failure within 28 days of enrollment. Treatment failure is defined as:

- Progression to WHO classification level 6 or greater including the need for high-flow oxygen or non-invasive ventilation
- Receiving salvage therapy with a non-study immune-modulator (Appendix A).
- Lost to follow-up through hospital transfer, within the 14-day primary treatment period.
- Discontinuation of study drug for any cause prior to day 14 or hospital discharge will be considered as a treatment failure, except for those for whom study drug was temporarily suspended due to a decrease in renal function (creatinine clearance of < 60 mL/min), other reasons for temporary cessation of treatment listed in Section 7.3.2 of the protocol, or for discontinuation in the case of pregnancy. These subjects will be followed for the primary endpoint at 28 days with long-term follow-up at day 56.

Subjects who complete 14 days of treatment but remain hospitalized but do not meet the criteria for treatment failure, will not considered be as treatment failures with respect to the primary endpoint.

# 8.2. Analysis of the Primary Efficacy Endpoint

The proportion of subjects in each treatment group who reach the study endpoint of treatment failure by 28 days will be compared to placebo using Fisher's Exact 2-sided test of proportions. Additionally, the frequency for each outcome (intubation, ECMO, death) will be determined within each group. The ITT, mITT and PP analysis populations will be used to analyze the primary endpoint.

# 8.3. Definition of the Exploratory Efficacy Endpoints

Exploratory endpoints include the following which will be summarized using the PP populations by treatment group received:

- Assess the number of days of hospitalization relative to treatment group
- Assess the number of days requiring ICU care relative to treatment group. If a subject does not require ICU care, the number of days will be set to zero for the group summary. The number of ICU days will be summarized for all subjects in each group and for the proportion of those who are actually in ICU.
- Assess the number of days of non-invasive or mechanical ventilation relative to treatment group. If a subject does not require non-invasive or mechanical ventilation, the number of days will be set to zero for the group summary. The number of mechanical ventilation


days will be summarized for all subjects in each group and for the proportion of those who are actually on mechanical ventilation.

- Assess incidence of WHO COVID-19 Classification levels relative to baseline serum IL-6 level
- Assess incidence of WHO COVID-19 Classification levels relative to baseline serum ferritin level
- Assess incidence of WHO COVID-19 Classification levels relative to baseline CRP
- Assess trough level of GLS-1027 relative to serum creatinine
- Assess the maximal level of Positive End-Expiratory Pressure (PEEP) for subjects who are intubated relative to treatment group.
- Assess the number of days of PEEP > 5 cm H2O for subjects who are intubated relative to treatment group
- Assessment of WHO COVID-19 Classification at 28 day relative to treatment group
- Assess SARS-CoV-2 IgM antibody responses relative to treatment group

No adjustments or imputations will be made for deaths or other forms of missingness except those already described above.

Corticosteroids will be recorded as a prior or concomitant medication. Subgroup analysis will be performed to compare outcomes relative to treatment group and relative to use or non-use of corticosteroids. Primary treatment outcomes will be determined from the time of enrollment through to Day 28.

# 8.4. Analysis of the Exploratory Efficacy Endpoints

PEEP values during intubation will be plotted separately by treatment over time. Assessment of WHO COVID-19 Classification at 28 day relative to treatment group is discussed in Sections 8.1 and 8.2. Shift tables for worst (most extreme) values of serum IL-6 level, serum ferritin level, and CRP relative to baseline will be presented for each WHO COVID-19 Classification level.

The number of days in ICU, requiring mechanical ventilation and of PEEP > 5 cm H<sub>2</sub>O will be summarized by treatment using descriptive statistics (sample size, mean, median, SD, minimum, maximum).

The number and percentage of subjects will be summarized by treatment according to their SARS-CoV-2 IgM antibody response. The above exploratory endpoint analyses will be presented for the PP population and individual results will be listed by treatment and study day. No formal statistical analysis is planned.


The relationship of trough level of GLS-1027 to serum creatinine relative to treatment group will be examined on an adhoc basis and is outside the scope of this document.

### 9. SAFETY ANALYSES

All safety analyses will be based on the Safety Population.

#### 9.1. Adverse Events

An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body, or worsening of a pre-existing condition, temporally associated with the use of a product whether or not considered related to the use of the product. In this study, such changes will be monitored, classified, and summarized, as Clinical or Laboratory AEs. Medical conditions/diseases present before starting the investigational drug will be considered adverse events only if they worsen after starting study treatment. Verbatim terms on CRFs will be mapped to preferred terms (PTs) and system organ classes (SOCs) using the Medical Dictionary for Regulatory Activities (MedDRA) (version 23.0).

# **9.1.1. Severity**

AEs are graded by the investigator as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (potentially life threatening) or Grade 5 (death) according to the NCI Common Terminology Criteria for Adverse Events version 5.0.

# 9.1.2. Relationship

Based on the criteria described below, AEs will be classified according to one of the following categories:

- Related the investigator considers that there is a causal relationship between the event and study drug
- Probably related the investigator considers that there is a probability of a causal relationship of the event to the study drug
- Possibly related the investigator considers that there is a possible causal relationship of the event to the study drug
- Unlikely related the investigator considers that there is an unlikely causal relationship of the event to the study drug
- Not related the investigator considers that the event has no relationship to administration of the study drug

For the purpose of analysis, related AEs are those reported as "Related," "Probably related," "Possibly related" and unrelated AEs are those reported as "Unlikely related" or "Not related." Events for which the investigator did not record relationship will be considered related for analysis. Data listings will show relationship as missing.

#### 9.1.3. Serious Adverse Events

An SAE is any AE that meets one of the following conditions:


- Is immediately life-threatening (e.g., participant was, in the view of the Investigator, at immediate risk of death from the event as it occurred);
- Requires or prolongs hospitalization;
- Results in congenital anomaly or birth defect;
- Results in persistent or significant disability/incapacity;
- Is an important medical event that may not result in death or be life threatening, but based upon appropriate medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed above;
- Results in death.

# 9.1.4. Treatment-Emergent Adverse Events (TEAEs)

# 9.1.4.1. Definition of Treatment-Emergent

TEAEs include the following:

- a) Post-treatment complications that occur as a result of protocol mandated procedure.
- b) Any pre-existing condition that increases in severity, or changes in nature during or as a consequence of the study drug phase of a human clinical trial, will also be considered an AE.
- c) Complications and termination of pregnancy; see protocol v5.0 section 7.1.7 for additional information.
- d) Non-elective medical or surgical procedures.

# 9.1.4.2. Incomplete Dates

If the date of onset is incomplete, then the month and year (or year alone if month is not recorded) of onset determine treatment emergence as follows. The event is treatment emergent if the month and year of onset (or year of onset) of the event is the same as or after the month and year (or year) of date of first dose.

#### 9.1.5. Summaries of Adverse Events

An overall summary of AEs will display, by treatment, the number and percentage of subjects who had any TEAE, whose strongest TEAE relationship to study drug is related or not related, whose maximum TEAE severity is mild, moderate, or severe, who had any SAE, any Serious TEAE, any TEAE leading to study discontinuation, and any TEAE leading to death.

The following summaries (number and percentage of subjects) of AEs (by SOC and PT) will be provided by treatment:

- All TEAEs
- All TEAEs by strongest relationship
- All TEAEs by maximum severity grade
- All Related TEAEs by maximum severity grade


- All Serious AEs
- All Serious TEAEs
- All TEAEs leading to study discontinuation
- All TEAEs leading to death

These summaries will present the number and percentage of subjects with at least one qualifying AE. Subjects may have more than one AE per SOC and PT. Each summary will be ordered by descending order of incidence of SOC and PT within each SOC.

In addition to the by-treatment summaries, data listings will be provided for the following:

- All AEs (with a flag indicating whether the event is treatment emergent)
- SAEs
- AEs leading to study discontinuation
- Deaths

# 9.2. Clinical Laboratory Evaluations

Continuous response variables per time point will be summarized with mean, median, minimum, and maximum values. Categorical response variables will be summarized per time point with percentages. Shift from baseline in laboratory parameter results (indicated as Low, Normal, or High) will be summarized for the worse (most extreme) post-baseline assessment. Mean (+/- SD) laboratory parameter values of interest will be graphically presented over time by treatment. All laboratory parameters will be listed and include indicators for low/high and clinical significance as determined by the investigator.

### 9.3. Vital Signs

Vital signs (temperature, heart rate, systolic blood pressure (SBP), diastolic blood pressure (DBP)) will be summarized using descriptive statistics (sample size, mean, SD, median, minimum, and maximum) at baseline and at each post-baseline time point by treatment. Change from baseline will also be summarized at each post-baseline time point. Mean (+/- SD) vital sign values will be graphically presented over time by treatment. All vital signs results will be listed.

# 9.4. ECG Results

Shift from baseline in 12-Lead ECG overall interpretation (results are Normal, Abnormal Not Clinically Significant (NCS), or Abnormal Clinically Significant (CS)) will be summarized at each post-baseline study day by treatment. Mean (+/- SD) continuous ECG parameter values will be graphically presented over time by treatment.

Additionally, the number and percentage of subjects will be summarized for the following QTcF Interval result categories at baseline and study day 15 by treatment:

- <=450 msec (males) or <=470 msec (females)
- >450 msec (males) or >470 msec (females)


- Change from baseline <=60 msec (only applies to post-baseline visits)
- Change from baseline >60 msec (only applies to post-baseline visits)

A listing of ECG results will present the interpretations of abnormalities and whether these are considered clinically significant by the investigator.

# 9.5. Physical Exam

Physical exam findings will be listed.

# 9.6. Urine Pregnancy Test

Pregnancy test results will be listed.

# 9.7. Other Data

Chest x-ray scores, nasal oxygen (O<sub>2</sub>) administration and flow rate, and CPAP usage and PEEP, % FiO2 if mechanically ventilated, ECMO treatment will be presented in listings. The number of days of nasal oxygen (O<sub>2</sub>) administration and flow rate, level of PEEP, % of FiO2 if mechanically ventilated, ECMO treatment and CPAP usage, will be summarized by treatment using descriptive statistics (sample size, mean, median, SD, minimum, maximum).


#### APPENDIX A: PRESENTATION OF DATA AND PROGRAMMING SPECIFICATIONS

#### **Tables**

- Formal organization of tabulations may be changed during programming if appropriate, e.g., tables for the different variables may be combined into a single table, or tables with more than one variable may be split into several tables.
- Means and medians will be presented to one more decimal place than the raw data. SDs will be presented to two more decimal places than the raw data. Minimums and maximums will be reported with the same number of decimal places as the raw data.
- Percentages will be presented to the tenths place.
- For frequency counts of categorical variables, categories whose counts are zero will be displayed for the sake of completeness. For example, if none of the subjects discontinue due to "lost to follow-up," this reason will be included in the table with a count of 0. Categories with zero counts will not have zero percentages displayed.
- The last footnote will be "Reference: xxx", where xxx indicates the source listing number(s).

# Listings

- Formal organization of the listing may be changed during programming if appropriate, e.g., additional variables may be included, change in the column order, or the listing may be split into multiple parts due to space constraints, etc.
- If not otherwise specified, all data listings will be sorted by treatment, subject number, visit, and date/time as appropriate.
- All date values will be presented in an ISO 8601 date (e.g., 2001-08-29) format.
- All observed time values will be presented using a 24-hour clock HH:MM:SS format (e.g., 01:35:45 or 11:26). Seconds will only be reported if they were measured as part of the study.

# Missing or incomplete dates, i.e., AEs and concomitant medications

The most conservative approach will be systematically considered. If the AE onset date is missing or incomplete, it is assumed to have occurred during the study treatment phase (i.e., considered a TEAE) except if the partial onset date or other data such as the stop date, indicates differently. Similarly, a medication with partial start and stop dates could be considered as a concomitant treatment.

The following algorithms will be applied to missing and incomplete start and stop dates:

### **Start Dates**

- If the day portion of the start date is missing, then the start date will be estimated to be equal to the date of IP administration, provided the start month and year are the same as IP administration and the stop date is either after IP administration or completely missing. Otherwise, the missing day portion will be estimated as '01'.
- If both the day and month portions of the start date are missing, then the start date will be estimated to be equal to the date of IP administration, provided the start year is the same as IP administration and the stop date is either after IP administration or completely


- missing. Otherwise, the event will be assumed to start on the first day of the given year, e.g., 2013-??-?? is estimated as 2013-01-01.
- If the start date is completely missing and the stop date is either after IP administration or completely missing, the start date will be estimated to be the day of IP administration. Otherwise, the start date will be estimated to be the first day of the same year as the stop date. All other non-AE and non-concomitant medication day calculations where only partial dates are available will be handled as follows: the first day of the month will be used in the calculations if the day part of a start date is missing while January 1 will be employed if both the month and day parts of a start date are missing.

# **Stop Dates**

- If only the day of resolution is unknown, the day will be assumed to be the last of the month, e.g., 2013-01-?? will be treated as 2013-01-31.
- If both the day and month of resolution are unknown, the event will be assumed to have ceased on the last day of the year, e.g., 2013-??-?? will be treated as 2013-12-31.
- If the stop date is completely missing or the event is continuing, the event will be assumed to be after IP administration and will be left as missing.

#### **Standard Calculations**

Variables requiring calculation will be derived using the following formulas:

- Days A duration expressed in days between two dates (start date and end date) is calculated using the formulas noted below:
- duration in days = end date start date + 1, where end date  $\ge$  treatment start date
- duration in days = end date start date, where end date < treatment start date
- Months A duration expressed in months is calculated as the number days divided by 365.25/12 (~30.4).
- Years A duration expressed in years between one date (date1) and another later date (date2) is calculated using the formula: duration in years = (date2-date1+1)/365.25
- Height Height entries made in inches (in) are converted to centimeters (cm) using the following formula: height (cm) = height (in)  $\times 2.54$
- Weight Weight entries made in pounds (lb.) are converted to kilograms (kg) using the following formula: weight (kg) = weight (lb.) / 2.2046
- Temperature Temperature entries in degrees Fahrenheit are converted to degrees centigrade using the following formula: temp (degrees centigrade) = 5/9 × [temp (degrees Fahrenheit) 32]


- Change from baseline Change from baseline will be calculated as: Change = post baseline value baseline value
- Percent change from baseline Change from baseline will be calculated as: percent change from baseline = post baseline value – baseline value / baseline value × 100


# APPENDIX B: TABLE OF CONTENTS FOR STATISTICAL TABLES AND LISTINGS

The following TFL numbering is completed according to ICH guidelines. The ICH heading number and description are in **bold**. Minor changes from this planned index do not need to be amended in the SAP. Formal organization of tabulations may be changed during programming if appropriate, e.g., tables for the different variables may be combined into a single table, or tables with more than one variable may be split into several tables.

# **List of Tables**

| ICH | Table | |
|---|---|---|
| Heading | Number | Table Description |
| 14.1 | | DEMOGRAPHIC/BASELINE DATA |
| | 14.1.1.1 | Subject Disposition (All Subjects) |
| | 14.1.1.2 | Reason for Screen Failure (All Screen Failure Subjects) |
| | 14.1.2 | Demographic and Baseline Characteristics (ITT Population) |
| | 14.1.3 | Medical History (ITT Population) |
| | 14.1.4 | Prior and Concomitant Medications (ITT Population) |
| | 14.1.5 | Treatment Exposure (Safety Population) |
| 14.2 | | EFFICACY DATA |
| | 14.2.1.1 | Analysis of Overall Treatment Failure (ITT Population) |
| | 14.2.1.2 | Analysis of Overall Treatment Failure (mITT Population) |
| | 14.2.1.2 | Analysis of Overall Treatment Failure (PP Population) |
| | 14.2.2.1.1 | Summary of the Number of Days Requiring ICU Care (ITT |
| | | Population) |
| | 14.2.2.1.2 | Summary of the Number of Days Requiring ICU Care (PP |
| | | Population) |
| | 14.2.2.2.1 | Summary of the Number of Days on Mechanical Ventilation (ITT Population) |
| | 14.2.2.2.2 | Summary of the Number of Days on Mechanical Ventilation (PP |
| | 1 112121212 | Population) |
| | 14.2.2.3.1 | Summary of Number of Days Requiring Nasal Oxygen (O <sub>2</sub> ) Administration (ITT Population) |
| | 14.2.2.3.2 | Summary of Number of Days Requiring Nasal Oxygen (O <sub>2</sub> ) Administration (PP Population) |
| | 14.2.2.4.1 | Summary of Number of Days Requiring CPAP Usage (ITT Population) |
| | 14.2.2.4.2 | Summary of Number of Days Requiring CPAP Usage (PP Population) |
| | 14.2.2.5.1 | Summary of Number of Days Requiring ECMO Administration (ITT Population) |
| | 14.2.2.5.2 | Summary of Number of Days Requiring ECMO Administration (PP Population) |
| | 14.2.2.6.1 | Summary of Number of Days with PEEP > 5cm H2O (ITT Population) |

| ICH | Table | |
|---|---|---|
| Heading | Number | Table Description |
| g | 14.2.2.6.2 | Summary of Number of Days with PEEP > 5cm H2O (PP |
| | | Population) |
| | 14.2.2.7.1 | Summary of Maximal Levels of PEEP values (ITT Population) |
| | 14.2.2.7.2 | Summary of Maximal Levels of PEEP values (PP Population) |
| | 14.2.2.8.1 | Summary of the Number of Days in Hospital (ITT Population) |
| | 14.2.2.8.2 | Summary of the Number of Days in Hospital (PP Population) |
| | 14.2.3.1 | Cumulative Incidence of SARS-CoV-2 IgM Antibody Response by |
| | | Study Day (PP Population) |
| | 14.2.4.1 | WHO COVID-19 Classification Levels Relative to Baseline Serum |
| | | Ferritin Level |
| | 14.2.4.2 | WHO COVID-19 Classification Levels Relative to Baseline Serum |
| | | IL-6 Level |
| | 14.2.4.3 | WHO COVID-19 Classification Levels Relative to Baseline CRP |
| 14.3 | | SAFETY DATA |
| 14.3.1 | | Displays of Adverse Events |
| | 14.3.1.1 | Overall Summary of Treatment-Emergent Adverse Events (Safety |
| | 11212 | Population) |
| | 14.3.1.2 | Treatment-Emergent Adverse Events by System Organ Class and |
| | 11212 | Preferred Term (Safety Population) |
| | 14.3.1.3 | Treatment-Emergent Adverse Events by System Organ Class, |
| | | Preferred Term, and Strongest Relationship to Study Drug (Safety Population) |
| | 14.3.1.4 | Treatment-Emergent Adverse Events by System Organ Class, |
| | | Preferred Term, and Maximum Severity Grade (Safety Population) |
| | 14.3.1.5 | Related Treatment-Emergent Adverse Events by System Organ |
| | | Class, Preferred Term, and Maximum Severity Grade (Safety |
| | | Population) |
| 14.3.2 | | Serious and Significant Adverse Events |
| | 14.3.2.1 | Serious Adverse Events by System Organ Class and Preferred Term (Safety Population) |
| | 14.3.2.2 | Serious Treatment-Emergent Adverse Events by System Organ |
| | | Class and Preferred Term (Safety Population) |
| | 14.3.2.3 | Treatment-Emergent Adverse Events Leading to Study |
| | | Discontinuation by System Organ Class and Preferred Term |
| | | (Safety Population) |
| | 14.3.2.4 | Treatment-Emergent Adverse Events Leading to Death by System |
| | | Organ Class and Preferred Term (Safety Population) |
| 14.3.4 | | Laboratory |
| | 14.3.4.1 | Hematology (Safety Population) |
| | 14.3.4.2 | Chemistry (Safety Population) |
| | 14.3.4.3 | Shift from Baseline in Hematology Results by Test (Safety |
| | | Population) |

| ICH | Table | |
|---|---|---|
| Heading | Number | Table Description |
| | 14.3.4.4 | Shift from Baseline in Chemistry Results by Test (Safety |
| | | Population) |
| | 14.3.4.5 | Observed and Change from Baseline in Vital Sign Results by Test |
| | | and Study Day (Safety Population) |
| | 14.3.4.6.1 | Shift from Baseline in 12-Lead ECG Overall Interpretation by |
| | | Study Day (Safety Population) |
| | 14.3.4.6.2 | Summary of QTcF Interval (msec) by Study Day and Result |
| | | Category (Safety Population) |

# **List of Figures**

| ICH | Figure | |
|---|---|---|
| Heading | Number | Figure Description |
| 14.2 | | Efficacy Data |
| | 14.2.2.1 | Line Plots of Mean (+/- SD) PEEP Results During Intubation by |
| | | Study Day (ITT Population) |
| | 14.2.2.2 | Line Plots of Mean (+/- SD) PEEP Results During Intubation by |
| | | Study Day (PP Population) |
| 14.3.4 | | Laboratory |
| | 14.3.4.1 | Line Plots of Mean (+/- SD) Vital Sign Results by Test and Study |
| | | Day (Safety Population) |
| | 14.3.4.2 | Line Plots of Mean (+/- SD) 12-Lead ECG Results by Test and |
| | | Study Day (Safety Population) |

# **List of Data Listings**

| Number | ICH Heading | Listing | |
|---|---|---|---|
| 16.2.1 Discontinued Subjects | | Number | Listing Description |
| 16.2.1 Subject Disposition | | | |
| 16.2.2 Protocol Deviations | 16.2.1 | | |
| 16.2.3 Protocol Deviations | | 16.2.1 | |
| 16.2.3 Subjects Excluded from the Safety Analysis 16.2.4 Demographic and Baseline Data 16.2.4.1 Demographic and Baseline Characteristics 16.2.4.2 Medical History 16.2.4.3 Prior and Concomitant Medications 16.2.5 Exposure and/or Drug Concentration Data 16.2.5.1 Treatment Exposure 16.2.5.2 Study Drug Administration 16.2.5.3 Pharmacokinetic Assessment 16.2.5.4 Blood Draw 16.2.6 Individual Efficacy Response Data 16.2.6.1 WHO Clinical Classification 16.2.6.2 Mechanical Ventilation 16.2.6.3 Nasal Oxygen (O2) Administration 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission 16.2.6.5 SARS-CoV-2 IgM Antibody Titer and Response 16.2.7.1 Adverse Events listings 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | 16.2.2 | | |
| 16.2.4 Demographic and Baseline Data 16.2.4.1 Demographic and Baseline Characteristics 16.2.4.2 Medical History 16.2.4.3 Prior and Concomitant Medications 16.2.5.1 Exposure and/or Drug Concentration Data 16.2.5.2 Study Drug Administration 16.2.5.3 Pharmacokinetic Assessment 16.2.5.4 Blood Draw 16.2.5.4 Blood Draw 16.2.6.1 WHO Clinical Classification 16.2.6.2 Mechanical Ventilation 16.2.6.3 Nasal Oxygen (O2) Administration 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission 16.2.6.5 SARS-CoV-2 IgM Antibody Titer and Response 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.2 | |
| 16.2.4 Demographic and Baseline Data 16.2.4.1 Demographic and Baseline Characteristics 16.2.4.2 Medical History 16.2.4.3 Prior and Concomitant Medications 16.2.5 Exposure and/or Drug Concentration Data 16.2.5.1 Treatment Exposure 16.2.5.2 Study Drug Administration 16.2.5.3 Pharmacokinetic Assessment 16.2.5.4 Blood Draw 16.2.6 Individual Efficacy Response Data 16.2.6.1 WHO Clinical Classification 16.2.6.2 Mechanical Ventilation 16.2.6.3 Nasal Oxygen (O2) Administration 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission 16.2.6.5 SARS-COV-2 IgM Antibody Titer and Response 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | 16.2.3 | | |
| 16.2.4.1 Demographic and Baseline Characteristics 16.2.4.2 Medical History 16.2.4.3 Prior and Concomitant Medications 16.2.5 Exposure and/or Drug Concentration Data 16.2.5.1 Treatment Exposure 16.2.5.2 Study Drug Administration 16.2.5.3 Pharmacokinetic Assessment 16.2.5.4 Blood Draw 16.2.6 Individual Efficacy Response Data 16.2.6.1 WHO Clinical Classification 16.2.6.2 Mechanical Ventilation 16.2.6.3 Nasal Oxygen (O2) Administration 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission 16.2.6.5 SARS-CoV-2 IgM Antibody Titer and Response 16.2.7 Adverse Events listings 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.8 Laboratory and Other Data 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.3 | |
| 16.2.4.2 Medical History 16.2.4.3 Prior and Concomitant Medications 16.2.5 Exposure and/or Drug Concentration Data 16.2.5.1 Treatment Exposure 16.2.5.2 Study Drug Administration 16.2.5.3 Pharmacokinetic Assessment 16.2.5.4 Blood Draw 16.2.6 Individual Efficacy Response Data 16.2.6.1 WHO Clinical Classification 16.2.6.2 Mechanical Ventilation 16.2.6.3 Nasal Oxygen (O2) Administration 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission 16.2.6.5 SARS-COV-2 IgM Antibody Titer and Response 16.2.7 Adverse Events 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.8 Laboratory and Other Data 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | 16.2.4 | | |
| 16.2.4.3 Prior and Concomitant Medications | | 16.2.4.1 | |
| 16.2.5 Exposure and/or Drug Concentration Data 16.2.5.1 Treatment Exposure 16.2.5.2 Study Drug Administration 16.2.5.3 Pharmacokinetic Assessment 16.2.5.4 Blood Draw 16.2.6 Individual Efficacy Response Data 16.2.6.1 WHO Clinical Classification 16.2.6.2 Mechanical Ventilation 16.2.6.3 Nasal Oxygen (O2) Administration 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission 16.2.6.5 SARS-CoV-2 IgM Antibody Titer and Response 16.2.7 Adverse Events listings 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.8 Laboratory and Other Data 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | | |
| 16.2.5.1 Treatment Exposure 16.2.5.2 Study Drug Administration 16.2.5.3 Pharmacokinetic Assessment 16.2.5.4 Blood Draw 16.2.6 Individual Efficacy Response Data 16.2.6.1 WHO Clinical Classification 16.2.6.2 Mechanical Ventilation 16.2.6.3 Nasal Oxygen (O2) Administration 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission 16.2.6.5 SARS-CoV-2 IgM Antibody Titer and Response 16.2.7 Adverse Events listings 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.7.4 Deaths 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.4.3 | Prior and Concomitant Medications |
| 16.2.5.2 Study Drug Administration 16.2.5.3 Pharmacokinetic Assessment 16.2.5.4 Blood Draw 16.2.6 Individual Efficacy Response Data 16.2.6.1 WHO Clinical Classification 16.2.6.2 Mechanical Ventilation 16.2.6.3 Nasal Oxygen (O2) Administration 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission 16.2.6.5 SARS-CoV-2 IgM Antibody Titer and Response 16.2.7 Adverse Events listings 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.7.4 Deaths 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | 16.2.5 | | Exposure and/or Drug Concentration Data |
| 16.2.5.3 Pharmacokinetic Assessment 16.2.5.4 Blood Draw 16.2.6 Individual Efficacy Response Data 16.2.6.1 WHO Clinical Classification 16.2.6.2 Mechanical Ventilation 16.2.6.3 Nasal Oxygen (O2) Administration 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission 16.2.6.5 SARS-CoV-2 IgM Antibody Titer and Response 16.2.7 Adverse Events listings 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.7.4 Deaths 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.5.1 | Treatment Exposure |
| 16.2.6 Individual Efficacy Response Data 16.2.6.1 WHO Clinical Classification 16.2.6.2 Mechanical Ventilation 16.2.6.3 Nasal Oxygen (O <sub>2</sub> ) Administration 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission 16.2.6.5 SARS-CoV-2 IgM Antibody Titer and Response 16.2.7 Adverse Events listings 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.7.4 Deaths 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.5.2 | |
| 16.2.6 Individual Efficacy Response Data 16.2.6.1 WHO Clinical Classification 16.2.6.2 Mechanical Ventilation 16.2.6.3 Nasal Oxygen (O <sub>2</sub> ) Administration 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission 16.2.6.5 SARS-CoV-2 IgM Antibody Titer and Response Adverse Events listings 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.7.4 Deaths 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | | Pharmacokinetic Assessment |
| 16.2.6.1 WHO Clinical Classification 16.2.6.2 Mechanical Ventilation 16.2.6.3 Nasal Oxygen (O <sub>2</sub> ) Administration 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission 16.2.6.5 SARS-CoV-2 IgM Antibody Titer and Response 16.2.7 Adverse Events listings 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.7.4 Deaths 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.5.4 | Blood Draw |
| 16.2.6.2 Mechanical Ventilation 16.2.6.3 Nasal Oxygen (O <sub>2</sub> ) Administration 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission 16.2.6.5 SARS-CoV-2 IgM Antibody Titer and Response 16.2.7 Adverse Events listings 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.7.4 Deaths 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | 16.2.6 | | Individual Efficacy Response Data |
| 16.2.6.3 Nasal Oxygen (O <sub>2</sub> ) Administration 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission 16.2.6.5 SARS-CoV-2 IgM Antibody Titer and Response 16.2.7 Adverse Events listings 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.7.4 Deaths 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.6.1 | WHO Clinical Classification |
| 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission 16.2.6.5 SARS-CoV-2 IgM Antibody Titer and Response 16.2.7 Adverse Events listings 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.7.4 Deaths 16.2.8 Laboratory and Other Data 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.6.2 | Mechanical Ventilation |
| 16.2.6.5 SARS-CoV-2 IgM Antibody Titer and Response 16.2.7 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.7.4 Deaths Laboratory and Other Data 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.6.3 | Nasal Oxygen (O <sub>2</sub> ) Administration |
| 16.2.7 Adverse Events listings 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.7.4 Deaths 16.2.8 Laboratory and Other Data 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.6.4 | CPAP Use, ECMO Prescription, ICU Admission |
| 16.2.7.1 Adverse Events 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.7.4 Deaths 16.2.8 Laboratory and Other Data 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.6.5 | SARS-CoV-2 IgM Antibody Titer and Response |
| 16.2.7.2 Serious Adverse Events 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.7.4 Deaths 16.2.8 Laboratory and Other Data 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | 16.2.7 | | Adverse Events listings |
| 16.2.7.3 Adverse Events Leading to Study Discontinuation 16.2.7.4 Deaths 16.2.8 Laboratory and Other Data 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.7.1 | Adverse Events |
| 16.2.8 Laboratory and Other Data 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.7.2 | Serious Adverse Events |
| 16.2.8 Laboratory and Other Data 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.7.3 | Adverse Events Leading to Study Discontinuation |
| 16.2.8.1 Hematology 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.7.4 | Deaths |
| 16.2.8.2 Chemistry 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | 16.2.8 | | Laboratory and Other Data |
| 16.2.8.3 Vital Signs 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.8.1 | Hematology |
| 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | 16.2.8.2 | Chemistry |
| 16.2.8.4 12-Lead Electrocardiogram 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | | |
| 16.2.8.5 Physical Examination 16.2.8.6 Urine Pregnancy Test | | | |
| 16.2.8.6 Urine Pregnancy Test | | | |
| | | | · · |
| | | 16.2.8.7 | |

**APPENDIX C: TABLE LAYOUTS** 

Table 14.1.1.1
Subject Disposition
(All Subjects)

| Subject Status | GLS-1027 | GLS-1027 | Placebo | 0verall |
|----------------------------|-----------|-----------|-----------|-----------|
| | 120 mg | 360 mg | | |
| Screened | | | | xx |
| Screen Failure | | | | XX |
| ITT Population [1] | XX | XX | XX | XX |
| mITT Population [2] | xx | xx | XX | xx |
| Safety Population [3] | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| PP Population [4] | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Completed the study | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Discontinued the study | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Reason for discontinuation | , , | , , | , , | , , |
| <reason #1=""></reason> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <reason #2=""></reason> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <reason #3=""></reason> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

Percentages are based on the ITT Population, unless otherwise noted.

Reference: Listing 16.2.1

<sup>[1]</sup> The Intent-to-treat (ITT) Population includes all randomized to treatment allocation.

<sup>[2]</sup> The modified intention to treatment (mITT) population includes all participants who are randomized to a treatment allocation, and who have received at least one dose of study drug.

<sup>[3]</sup> The Safety Population includes all subjects in the ITT population who received at least one dose of study drug.

<sup>[4]</sup> The PP Population includes all safety subjects who complete the trial by meeting the endpoint or being discharged within 14 days without meeting the endpoint.

GeneOne Life Science Inc.

Page 1 of 1

Protocol: GLS27-005

Table 14.1.1.2
Reason for Screen Failure
(All Screen Failure Subjects)

| Reason | Overall<br>(xx) |
|-------------------------|-----------------|
| <reason #1=""></reason> | x (xx.x%) |
| <reason #2=""></reason> | x (xx.x%) |
| <reason #3=""></reason> | x (xx.x%) |

Reference: Listing 16.2.3

Table 14.1.2

Demographic and Baseline Characteristics
(ITT Population)

| Characteristic | GLS-1027 | GLS-1027 | | |
|---|---|---|---|---|
| | 120 mg | 360 mg | Placebo | Overall |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Age (years) | | | | |
| n | xx | XX | xx | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x | xx.x |
| Min, Max | XX, XX | xx, xx | XX, XX | xx, xx |
| <65 years | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| >=65 years | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Sex | | | | |
| Male | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Female | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Race | | | | |
| American Indian or Alaskan Native | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Asian | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Black or African American | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Native Hawaiian or Other Pacific Islander | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| White | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Other | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Ethnicity | | | | |
| Hispanic or Latino | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Not Hispanic or Latino | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Not Reported | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Unknown | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

Baseline is the last non-missing value prior to first dose of study treatment. Reference: Listing 16.2.4.1

Table 14.1.2

Demographic and Baseline Characteristics
(ITT Population)

| Characteristic | GLS-1027 | GLS-1027 | | |
|----------------|-------------|-------------|-------------|-------------|
| | 120 mg | 360 mg | Placebo | Overall |
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Height (cm) | | | | |
| n | XX | XX | XX | xx |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | xx.x | xx.x | xx.x | xx.x |
| Min, Max | XX, XX | XX, XX | xx, xx | xx, xx |
| leight (kg) | | | | |
| n | xx | XX | xx | XX |
| Mean (SD) | xx.x (x.xx) | xx.x(x.xx) | xx.x(x.xx) | xx.x(x.xx) |
| Median | xx.x | xx.x | xx.x | xx.x |
| Min, Max | XX, XX | XX, XX | xx, xx | xx, xx |
| BMI (kg/m^2) | | | | |
| n | XX | xx | xx | xx |
| Mean (SD) | xx.x (x.xx) | xx.x(x.xx) | xx.x(x.xx) | xx.x(x.xx) |
| Median | xx.x | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | XX, XX | xx, xx | xx, xx |

BMI = Body Mass Index

Baseline is the last non-missing value prior to first dose of study treatment. Note: Body mass index (BMI) calculated as weight (kg) / [[height (cm)/100]<sup>2</sup>]. Reference: Listing 16.2.4.1

Table 14.1.3 Medical History (ITT Population)

| System Organ Class<br>Preferred Term | GLS-1027<br>120 mg<br>(N=XX) | GLS-1027<br>360 mg<br>(N=XX) | Placebo<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| Subjects with at least one medical history event | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <pre><system #1="" class="" organ=""></system></pre> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <pre><preferred #1="" term=""></preferred></pre> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| System Organ Class #2> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| • | | | | |
| • | | | | |

MedDRA = Medical Dictionary for Regulatory Activities.

Medical history terms are coded using MedDRA version 23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC. At each level of summation (overall, SOC, PT), subjects reporting more than one medical history term are counted only once. Reference: Listing 16.2.4.2

GeneOne Life Science Inc.


Protocol: GLS27-005

Table 14.1.4
Prior and Concomitant Medications
(ITT Population)

| ATC Class | GLS-1027 | GLS-1027 | Placebo |
|---|---|---|---|
| Preferred Name | 120 mg | 360 mg | (N=XX) |
| | (N=XX) | (N=XX) | |
| Subjects who received any prior or concomitant | | | |
| medications | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Subjects who received any prior or concomitant corticosteroids | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| ATC Class # 1> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" name=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" name=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #3="" name=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <atc #="" 2="" class=""></atc> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" name=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" name=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #3="" name=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| • | , , | . , | , , |
| • | | | |

A concomitant medication is any medication that was ongoing or started on or after the date of first dose. A prior medication is defined as a medication that was administered up to 4 months prior to time of enrollment.

Medications are coded using WHODrug Global (March 2020) and ordered by descending order of overall incidence of ATC class and overall incidence of preferred name within each class. At each level of summation (overall, ATC class, preferred name), subjects reporting more than one medication are counted only once.

Reference: Listing 16.2.4.3

Programming Note: Sort table by descending overall count of ATC class and descending overall count of preferred name within each class.

Table 14.1.5
Treatment Exposure

| | (Cafaty Danulation) | | |
|---|---|---|---|
| | (Safety Population) | CLC 1027 | |
| | GLS-1027 | GLS-1027 | |
| | 120 mg | 360 mg<br>(N=XX) | Placebo<br>(N=XX) |
| | (N=XX) | | |
| Duration of exposure (days) [1] | | | |
| n | XX | xx | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | XX, XX | XX, XX |
| Total number of doses taken | | | |
| n | XX | xx | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx |
| Total number of doses missed | | | |
| n | XX | xx | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| Min, Max | xx, xx | xx, xx | XX, XX |

<sup>[1]</sup> Duration of exposure is defined as the date of last dose minus the date of first dose + 1. Reference: Listing 16.2.5.1.

Table 14.2.1.1

Analysis of Overall Treatment Failure
(ITT Population)

Overall/Subjects with prior or concomitant corticosteroids/Subjects without prior or concomitant corticosteroids

| | GLS-1027 | GLS-1027 | Placebo<br>(N=XX) |
|---|---|---|---|
| | 120 mg | 360 mg | |
| | (N=XX) | (N=XX) | |
| Treatment Failure [1] | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Achieved WHO level >=6 | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Lost to follow-up | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Withdrawal of informed consent | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Required salvage therapy | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Discontinued study drug prior to discharge | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Had missing assessment of WHO level classification | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| p-value [2] | 0.xxxx | 0.xxxx | , , |
| Maximum WHO Level = 6 (Intubation or Mechanical Ventilation) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Maximum WHO Level = 7 (Requirement for ECMO) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Maximum WHO Level = 8 (Death) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

<sup>[1]</sup> Subjects who met any of the reasons listed are considered treatment failures. Subjects who failed treatment for multiple reasons are counted once for each reason.

Reference: Listing 16.2.6.1

Programming note: Repeat for Table 14.2.1.2 Analysis of Overall Treatment Failure (mITT Population).

Programming note: Repeat for Table 14.2.1.3 Analysis of Overall Treatment Failure (PP Population).

Programming note: P-values will not be provided for corticosteroid use/non-use subset pages.

<sup>[2]</sup> P-value is calculated using a Fisher's exact test and compares the active treatment to placebo. Will only be provided for the 120 mg group if the 360 mg group is significant.

GeneOne Life Science Inc.

Page 1 of 1

Protocol: GLS27-005

Table 14.2.2.1.1

Summary of the Number of Days Requiring ICU Care
(ITT Population)

| | GLS-1027 | GLS-1027 | Placebo |
|---|---|---|---|
| | 120 mg | 360 mg | (N=XX) |
| | (N=XX) | (N=XX) | , , |
| umber of Days Requiring ICU Care | | | |
| n | X | X | Х |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | x.xx | x.xx | x.xx |
| Hearan | | | xx.x, xx.x |

Reference: Listing xxxxx

Programming note: Repeat for Table 14.2.2.1.2 Summary of the Number of Days Requiring ICU Care (PP Population).
Protocol: GLS27-005

Table 14.2.2.2.1

Summary of the Number of Days on Mechanical Ventilation
(ITT Population)

| | GLS-1027 | GLS-1027 | Placebo |
|---|---|---|---|
| | 120 mg | 360 mg | (N=XX) |
| | (N=XX) | (N=XX) | , , |
| umber of Days on Mechanical Ventilation | | | |
| umber of Days on Mechanical Ventilation<br>n | х | x | × |
| | x<br>xx.xx (xx.xxx) | x<br>xx.xx (xx.xxx) | x<br>xx.xx (xx.xxx) |
| n | | | |

Reference: Listing 16.2.6.2

Programming note: Repeat for Table 14.2.2.2.2 Summary of the Number of Days on Mechanical Ventilation (PP Population).

Protocol: GLS27-005

Table 14.2.2.3.1 Summary of the Number of Days Requiring Nasal Oxygen  $(O_2)$  Administration (ITT Population)

| | GLS-1027 | GLS-1027 | Placebo |
|---|---|---|---|
| | 120 mg | 360 mg | (N=XX) |
| | (N=XX) | (N=XX) | |
| umber of Days Requiring Nasal Oxygen (O2) | | | |
| umber of Days Requiring Nasal Oxygen $(O_2)$ | x | x | x |
| | x<br>xx.xx (xx.xxx) | x<br>xx.xx (xx.xxx) | x<br>xx.xx (xx.xxx) |
| n | | | |

Reference: Listing 16.2.6.3

Programming note: Repeat for Table 14.2.2.3.2 Summary of the Number of Days Requiring Nasal Oxygen (O2) Administration (PP Population).

Protocol: GLS27-005

## Table 14.2.2.4.1 Summary of the Number of Days Requiring CPAP Usage (ITT Population)

| | GLS-1027 | GLS-1027 | Placebo |
|---|---|---|---|
| | 120 mg | 360 mg | (N=XX) |
| | (N=XX) | (N=XX) | , , |
| umber of Days Requiring CPAP Usage | | | |
| n | X | X | Х |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| | x.xx | x.xx | x.xx |
| Median | | | |

Reference: Listing 16.2.6.4

Programming note: Repeat for Table 14.2.2.4.2 Summary of the Number of Days Requiring CPAP Usage (PP Population).

Protocol: GLS27-005

Table 14.2.2.5.1

Summary of the Number of Days Requiring ECMO Administration (ITT Population)

| | GLS-1027 | GLS-1027 | Placebo |
|---|---|---|---|
| | 120 mg | 360 mg | (N=XX) |
| | (N=XX) | (N=XX) | |
| umber of Days Requiring FCMO Administration | | | |
| | x | × | × |
| n | x<br>xx.xx (xx.xxx) | x<br>xx.xx (xx.xxx) | x<br>xx.xx (xx.xxx) |
| umber of Days Requiring ECMO Administration<br>n<br>Mean (SD)<br>Median | | | x<br>xx.xx (xx.xxx)<br>x.xx |

Reference: Listing 16.2.6.5

Programming note: Repeat for Table 14.2.2.5.2 Summary of the Number of Days Requiring ECMO Administration (PP Population).

Protocol: GLS27-005

Table 14.2.2.6.1

Summary of the Number of Days with PEEP > 5 cm H20

(ITT Population)

| | GLS-1027 | GLS-1027 | Placebo |
|---|---|---|---|
| | 120 mg | 360 mg | (N=XX) |
| | (N=XX) | (N=XX) | , , |
| umber of Days with PEEP $>$ 5 cm $H_2O$ | | | |
| | V | X | X |
| n | X | ^ | ^ |
| | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| n<br>Mean (SD)<br>Median | | | |

Note: Only subjects who were intubated are included in this endpoint analysis.

Reference: Listing 16.2.6.2

Programming note: Repeat for Table 14.2.2.6.2 Summary of the Number of Days with PEEP > 5 cm H2O (PP Population).

Protocol: GLS27-005

## Table 14.2.2.7.1 Summary of Maximal Levels of PEEP Values (ITT Population)

| | GLS-1027 | GLS-1027 | Placebo |
|----------------------|----------------|----------------|----------------|
| | 120 mg | 360 mg | (N=XX) |
| | (N=XX) | (N=XX) | |
| aximal Level of PEEP | | | |
| n | X | x | Х |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | x.xx | x.xx | x.xx |
| Min, Max | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x |

Note: Only subjects who were intubated are included in this endpoint analysis.

Reference: Listing 16.2.6.2

Programming note: Repeat for Table 14.2.2.7.2 Summary of Maximal Levels of PEEP Values (PP Population).

Protocol: GLS27-005

Table 14.2.2.8.1
Summary of the Number of Days in Hospital
(ITT Population)

| | GLS-1027 | GLS-1027 | Placebo |
|---------------------------|----------------|----------------|----------------|
| | 120 mg | 360 mg | (N=XX) |
| | (N=XX) | (N=XX) | · · · |
| umber of Days in Hospital | | | |
| n | X | x | x |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | x.xx | x.xx | x.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |

Reference: Listing xxxxx

Programming note: Repeat for Table 14.2.2.8.2 Summary of the Number of Days in Hospital (PP Population).

Table 14.2.3.1

Cumulative Incidence of SARS-CoV-2 IgM Antibody Response by Study Day

(PP Population)

| Study Day | GLS-1027 | GLS-1027 | Placebo |
|-----------|-----------|-----------|-----------|
| Responded | 120 mg | 120 mg | (N=XX) |
| | (N=XX) | (N=XX) | `n(%)´ |
| | , | , | |
| Day 1 | | | |
| n | X | X | X |
| Yes | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| No | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 2 | | | |
| n | X | x | Х |
| Yes | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| No | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 3 | | | |
| n | X | X | X |
| Yes | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| No | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 4 | | | |
| n | X | X | X |
| Yes | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| No | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | (, | ~ () | . (, |
| •• | | | |

The incidence of antibody response is summarized based on results obtained at or prior to the study day. Reference: Listing 16.2.6.3

Table 14.2.4.1
WHO COVID-19 Classification Levels Relative to Baseline Serum Ferritin Level
(PP Population)

| | | | GL | S-1027 | | | GLS-1027 | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | L20 mg | | | 360 mg | | | Placebo | | | 0verall | |
| WHO Classification | (N=XX) | | | | | | (N=XX) | | | (N=XX) | | (N=XX) | | |
| Level | Serum Ferritin [1] | Post-Baseline | | | | | Post-Baseline | | | Post-Baseline | | | Post-Baseline | |
| | Baseline | Low | N | lormal | High | Low | Normal | High | Low | Normal | High | Low | Normal | High |
| 5 | n | х | | х | x | x | х | х | х | х | x | x | х | х |
| | Low | | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx | .x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.) |
| | Normal | | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx | .x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| | High | | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx | .x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| 6 | n | х | | х | x | x | х | х | х | х | x | x | х | х |
| | Low | | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx | .x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| | Normal | | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx | .x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| | High | | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx | .x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| 7 | n | х | | х | x | x | х | х | х | х | x | x | х | х |
| | Low | | | | | XX | XX | XX | XX | XX | XX | XX | xx | XX |
| | | xx (xx | .x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| | Normal | | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx | .x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| | High | | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx | .x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| 8 | n | х | | х | x | x | x | х | х | х | x | х | x | х |
| | Low | | | | | XX | XX | XX | XX | XX | XX | XX | XX | xx |
| | | xx (xx | .x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| | Normal | | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx | .x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| | High | | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx | .x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |

<sup>[1]</sup> Worst (most extreme) values presented for serum ferritin.

Reference: Listing xx.x.x.x

date time

Table 14.2.4.2 WHO COVID-19 Classification Levels Relative to Baseline Serum IL-6 Level (PP Population)

| | | | GL | .S-1027 | | | GLS-1027 | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | .20 mg | | | 360 mg | | | Placebo | | | Overall | |
| WHO Classification | | (N=XX) | | | | | (N=XX) | | | (N=XX) | | | (N=XX) | |
| Level | Serum IL-6 [1] | | Post-Baseline | | | | Post-Baseline | | | Post-Baseline | | | Post-Baseline | |
| | Baseline | L | .ow N | lormal | High | Low | Normal | High | Low | Normal | High | Low | Normal | High |
| 5 | n | | x | x | x | x | x | x | x | x | x | x | x | х |
| | Low | | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx ( | xx.x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.) |
| | Normal | | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx ( | xx.x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.) |
| | High | | | | | XX | XX | XX | XX | XX | XX | XX | xx | XX |
| | | xx ( | xx.x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| 6 | n | | x | x | x | x | x | x | x | х | x | x | х | х |
| | Low | | | | | XX | xx | XX | XX | XX | XX | XX | xx | XX |
| | | xx ( | xx.x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| Norm | Normal | , | • | ` , | ` , | XX | xx | XX | XX | XX | XX | XX | xx | ` xx |
| | | xx ( | xx.x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| | High | ` | , | ` , | , , | XX | `xx´ | XX | XX | XX | XX | XX | `xx´ | ` xx |
| | G | xx ( | xx.x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| 7 | n | | x | x | x | x | x | x | х | х | x | х | х | х |
| | Low | | | | | XX | xx | XX | XX | XX | XX | XX | xx | xx |
| | | xx ( | xx.x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| | Normal | , | • | | , , | XX | xx | XX | XX | XX | XX | XX | xx | · xx |
| | | xx ( | xx.x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| | High | , | • | | , , | XX | xx | XX | XX | XX | XX | XX | xx | · xx |
| | J | xx ( | xx.x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| 8 | n | | x | x | × | х | x | x | x | x | x | x | x | x |
| | Low | | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx ( | xx.x) xx | (xx.x)xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| | Normal | , | • | • | | xx | xx | XX | XX | XX | xx | XX | XX | · xx |
| | | xx ( | xx.x) xx | (xx.x) xx | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |
| | High | , | • | • | . , | xx | xx | xx | xx | xx | xx | xx | xx | ` xx |
| | Ŭ | xx ( | xx.x)xx | (xx.x) xx | ( ( x x ) | (xx x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx. |

<sup>[1]</sup> Worst (most extreme) values presented for serum IL-6. Reference: Listing xx.x.x.x

date time

Table 14.2.4.3 WHO COVID-19 Classification Levels Relative to Baseline CRP (PP Population)

| | | | GLS-1027 | | | GLS-1027 | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 120 mg | | | 360 mg | | | Placebo | | | Overall | |
| WHO Classification | 600 [4] | (N=XX) | | | | (N=XX) | | | (N=XX) | | (N=XX)<br>Post-Baseline | | |
| Level | CRP [1] | | Post-Baseline | | | | Post-Baseline | | | Post-Baseline | | | |
| | Baseline | Low | Normal | High | Low | Normal | High | Low | Normal | High | Low | Normal | High |
| 5 | n | х | х | x | x | х | х | x | x | х | х | х | х |
| | Low | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx.x | ) xx (xx.x) x | x (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.) |
| | Normal | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx.x | ) xx (xx.x) x | x (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.) |
| | High | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx.x | ) xx (xx.x) x | x (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.) |
| 6 | n | х | х | x | х | x | x | x | x | х | х | x | х |
| | Low | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx.x | ) xx (xx.x) x | x (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.) |
| | Normal | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx.x | ) xx (xx.x) x | x (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.) |
| | High | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx.x | ) xx (xx.x) x | x (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.) |
| 7 | n | х | X | x | x | x | x | x | x | х | х | x | х |
| | Low | | | | XX | XX | XX | XX | XX | XX | XX | XX | xx |
| | | xx (xx.x | ) xx (xx.x) x | x (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.) |
| | Normal | | | | XX | xx | XX | XX | XX | XX | XX | xx | XX |
| | | xx (xx.x | ) xx (xx.x) x | x (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.) |
| | High | | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx.x | ) xx (xx.x) x | x (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.) |
| 8 | n | x | x | х | x | x | x | x | x | x | x | x | х |
| | Low | | | | XX | XX | XX | XX | XX | XX | XX | XX | xx |
| | | xx (xx.x | ) xx (xx.x) x | x (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.) |
| | Normal | • | • | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | xx (xx.x | ) xx (xx.x) x | x (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.) |
| | High | • | | • | xx | XX | XX | xx | xx | XX | XX | XX | · xx |
| | - | xx (xx.x | ) xx (xx.x) x | x (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.) |

<sup>[1]</sup> Worst (most extreme) values presented for CRP. Reference: Listing xx.x.x.x

date time

Table 14.3.1.1

Overall Summary of Treatment-Emergent Adverse Events
(Safety Population)

| | GLS-1027 | GLS-1027 | Placebo | Overall |
|---|---|---|---|---|
| | 120 mg | 360 mg | (N=XX) | (N=XX) |
| | (N=XX) | (N=XX) | | |
| ubjects with any TEAE | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| ubjects whose strongest TEAE relationship to study drug is | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| ubjects whose strongest TEAE relationship to study drug is out related [2] | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| ubjects whose maximum TEAE severity grade is grade 1 [3] | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| ubjects whose maximum TEAE severity grade is grade 2 [3] | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| ubjects whose maximum TEAE severity grade is grade 3 [3] | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| ubjects whose maximum TEAE severity grade is grade 4 [3] | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| ubjects with any SAE | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| ubjects with any Serious TEAE | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| ubjects with any TEAE leading to study discontinuation | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| ubjects with any TEAE leading to death | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

AE = Adverse Event; SAE = Serious Adverse Event; TEAE = Treatment-Emergent Adverse Event;

<sup>[1]</sup> Related TEAEs are those with a relationship of related, possibly related, or probably related. If the relationship is missing, it is considered related.

<sup>[2]</sup> Not related TEAEs are those with a relationship of unlikely related or not related.

<sup>[3]</sup> Severity grades are determined according to the NCI Common Terminology Criteria for Adverse Events version 5.0. Reference: Listing 16.2.7.1

Table 14.3.1.2

Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)

| System Organ Class | GLS-1027 | GLS-1027 | Placebo | Overall |
|---|---|---|---|---|
| Preferred Term | 120 mg | 360 mg | (N=XX) | (N=XX) |
| | (N=XX) | (N=XX) | | |
| Subjects with at least | | | | |
| one TEAE | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <system #1="" class="" organ=""></system> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <system #2="" class="" organ=""></system> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| • | | | | |
| • | | | | |

AE=Adverse Event; TEAE = Treatment-Emergent Adverse Event; MedDRA = Medical Dictionary for Regulatory Activities.

AEs are coded using MedDRA version 23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC. At each level of summation (overall, SOC, PT), subjects reporting more than one TEAE are counted only once.

Reference: Listing 16.2.7.1

Table 14.3.1.3

Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Strongest Relationship to Study Drug
(Safety Population)

| System Organ Class Preferred Term | | -1027<br>0 mg | GLS-1027<br>360 mg | | | icebo<br>I=XX) | Overall<br>(N=XX) | |
|---|---|---|---|---|---|---|---|---|
| | (N=XX) | | (N=XX) | | · | • | | |
| | Related | Not Related | Related | Not Related | Related | Not Related | Related | Not Related |
| Subjects with at least one related TEAE | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <system #1="" class="" organ=""></system> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <system #2="" class="" organ=""></system> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| • | | | | | | | | |

AE=Adverse Event; TEAE = Treatment-Emergent Adverse Event; MedDRA = Medical Dictionary for Regulatory Activities.

AEs are coded using MedDRA version 23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC. At each level of summation (overall, SOC, PT), subjects reporting more than one TEAE are counted only once using the strongest relationship. Related TEAEs are those with a relationship of related, possibly related, or probably related. If the relationship is missing, it is considered related. Not Related TEAEs are those with a relationship of unlikely related or not related. Reference: Listing 16.2.7.1


GeneOne Life Science Inc. Protocol: GLS27-005

Table 14.3.1.4

Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Severity Grade
(Safety Population)

| System Organ Class | | | | |
|---|---|---|---|---|
| Preferred Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Subjects with at least one TEAE | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <system #1="" class="" organ=""></system> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <system #2="" class="" organ=""></system> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

AE=Adverse Event; TEAE = Treatment-Emergent Adverse Event; MedDRA = Medical Dictionary for Regulatory Activities

AEs are coded using MedDRA version 23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC.

At each level of summation (overall, SOC, PT), subjects reporting more than one TEAE are counted only once using the highest grade.

Severity grades are determined according to the NCI Common Terminology Criteria for Adverse Events version 5.0.

Reference: Listing 16.2.7.1

## Repeat Table Layout for:

Table 14.3.1.5

Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Severity Grade (Safety Population)

Table 14.3.2.1 Serious Adverse Events by System Organ Class and Preferred Term (Safety Population)

| System Organ Class<br>Preferred Term | GLS-1027<br>120 mg<br>(N=XX) | GLS-1027<br>360 mg<br>(N=XX) | Placebo<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| Subjects with at least one serious AE | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <system #1="" class="" organ=""></system> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| System Organ Class #2> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <pre><preferred #1="" term=""></preferred></pre> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| • | | | | |

AE=Adverse Event; Adverse Event; MedDRA = Medical Dictionary for Regulatory Activities.

AEs are coded using MedDRA v23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC. At each level of summation (overall, SOC, PT), subjects reporting more than one AE are counted only once. Reference: Listing 16.2.7.2

date time

Table 14.3.2.2

Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)

| System Organ Class<br>Preferred Term | GLS-1027<br>120 mg<br>(N=XX) | GLS-1027<br>360 mg<br>(N=XX) | Placebo<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| Subjects with at least one serious TEAE | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <system #1="" class="" organ=""></system> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <pre><preferred #1="" term=""></preferred></pre> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| :System Organ Class #2> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <pre><preferred #1="" term=""></preferred></pre> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| • | , , | | . , | , , |

AE=Adverse Event; TEAE = Treatment-Emergent Adverse Event; MedDRA = Medical Dictionary for Regulatory Activities.

AEs are coded using MedDRA v23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC. At each level of summation (overall, SOC, PT), subjects reporting more than one TEAE are counted only once.

Reference: Listing 16.2.7.2

Table 14.3.2.3

Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term
(Safety Population)

| System Organ Class<br>Preferred Term | GLS-1027<br>120 mg | GLS-1027<br>360 mg | Placebo<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| | (N=XX) | (N=XX) | | |
| Subjects with at least one TEAE leading to study | | | | |
| discontinuation | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <system #1="" class="" organ=""></system> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| System Organ Class #2> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <pre><preferred #1="" term=""></preferred></pre> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| • | | | | |

AE=Adverse Event; TEAE = Treatment-Emergent Adverse Event; MedDRA = Medical Dictionary for Regulatory Activities

AEs are coded using MedDRA v23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC. At each level of summation (overall, SOC, PT), subjects reporting more than one TEAE are counted only once.

Reference: Listing 16.2.7.4

Table 14.3.2.4

Treatment-Emergent Adverse Events Leading to Death by System Organ Class and Preferred Term
(Safety Population)

| System Organ Class<br>Preferred Term | GLS-1027<br>120 mg<br>(N=XX) | GLS-1027<br>360 mg<br>(N=XX) | Placebo<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| Subjects with at least one TEAE leading to death | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <system #1="" class="" organ=""></system> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| :System Organ Class #2> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| • | | | | |

AE = Adverse Event; TEAE = Treatment-Emergent Adverse Event; MedDRA = Medical Dictionary for Regulatory Activities

AEs are coded using MedDRA v23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC. At each level of summation (overall, SOC, PT), subjects reporting more than one TEAE are counted only once.

Reference: Listing 16.2.7.1

Table 14.3.4.1 Hematology (Safety Population)

| | | GLS- | 1027 | GLS- | 1027 | Plac | cebo | To- | tal |
|---|---|---|---|---|---|---|---|---|---|
| | | | ) mg | 366 | ) mg | ( N= | xx) | | : xx) |
| Test | Time Point | (N=xx) | | | ·xx) | ` | , | • | • |
| | | Result | Change from<br>Baseline | Result | Change from<br>Baseline | Result | Change from<br>Baseline | Result | Change from<br>Baseline |
| <test #1<br="">(<unit>)</unit></test> | > Baseline | | | | | | | | |
| | n | XX | | xx | | xx | | XX | |
| | Mean (SD) | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | | xx.x (xx.xx) | |
| | Median | xx.x | | XX.X | | XX.X | | XX.X | |
| | Min, Max | XX, XX | | xx, xx | | xx, xx | | xx, xx | |
| | Day 2 | | | | | | | | |
| | n | xx | XX | XX | XX | XX | XX | XX | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | xx.x | XX.X | XX.X | xx.x | xx.x | xx.x |
| | Min, Max | XX, XX | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| | Etc. | | | | | | | | |

Baseline is the last non-missing value prior to first dose of study treatment.

Reference: Listing 16.2.8.1

Programming Note: Continue for all hematology tests.

Repeat Table 14.3.4.1 Layout for:

Table 14.3.4.2 Chemistry (Safety Population) Protocol: GLS27-005

Table 14.3.4.3
Shift from Baseline in Hematology Results by Test
(Safety Population)

| 「est [1] | | GLS-1027 | | | GLS-1027 | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 120 mg | | 360 mg | | | Place | bo | | 0verall | |
| | (N=XX)<br>Baseline | | | | (N=XX) | | | (N=XX) | | | (N=XX)<br>Baseline | |
| | | | | Baseline | | | Baseline | | | | | |
| <del>-</del> | Low | Normal | High | Low | Normal | High | Low | Normal | High | Low | Normal | High |

xx (xx.x) xx (xx

xx (xx.x) xx (

xx (xx.x) xx (xx

n

Low

Normal High

Baseline is the last non-missing value prior to first dose of study treatment.

Percentages are based on n, the number of subjects with both a baseline and post-baseline result at the study day.

Shifts are based on local labs from each site.

Reference: Listing 16.2.8.1

Programming Note: Continue for all hematology tests.

Repeat Table 14.3.4.1 Layout for:

Table 14.3.4.4

Shift from Baseline in Chemistry Results by Test and Study Day (Safety Population)

<sup>[1]</sup> Worst (most extreme) values presented for each test.

Table 14.3.4.5

Observed and Change from Baseline in Vital Sign Results by Test and Study Day
(Safety Population)

| Test | 0 | GLS-1027 GLS-1027 | | Placebo | | 0veral1 | | |
|---|---|---|---|---|---|---|---|---|
| Study Day | | 120 mg | | 360 mg | (N=) | (X) | (N= | XX) |
| | | (N=XX) | | (N=XX) | | | | |
| | Observed | Change from Baselin | e Observed | Change from Baseline | Change from | n Baseline | Change fro | m Baseline |
| <test #1=""> (units)</test> | ) | | | | | | | |
| Baseline ` | , | | | | | | | |
| n | X | | X | | X | | X | |
| Mean (SD) | xx.xx (xx.xxx) | | xx.xx (xx.xxx) | | xx.xx (xx.xxx) | | xx.xx (xx.xxx) | |
| Median | x.xx | | x.xx | | x.xx | | x.xx | |
| Min, Max | xx.x, xx.x | | xx.x, xx.x | | xx.x, xx.x | | xx.x, xx.x | |
| Day 2 | | | | | | | | |
| 'n | X | × | X | × | X | x | X | X |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx | (xx.xx) | xx.xx (xx.xxx) |
| Median | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Day 3 | | | | | | | | |
| n | X | × | X | × | X | x | X | X |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | | | (xx.xx) | xx.xx (xx.xxx) |
| Median | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |

Baseline is the last non-missing value prior to first dose of study treatment.

Reference: Listing 16.2.8.3

date time

Programming Note: Continue for all vital sign tests.

Table 14.3.4.6.1 Shift from Baseline in 12-Lead ECG Overall Interpretation by Study Day (Safety Population)

| Study Day | | GLS-1027 | 1 | | GLS-102 | | | Placebo | ) | | 0verall | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 120 mg | | | 360 mg | • | | (N=XX) | | | (N=XX) | |
| | | (N=XX) | | | (N=XX) | • | | Baselin | e | | Baseline | |
| | | Baseline | ! | | Baseli | ne | | | | | | |
| | Normal | Abnormal NCS | SAbnormal CS | Normal | Abnormal N | NCS Abnormal CS | Normal | Abnormal N | CSAbnormal CS | Normal | Abnormal | Abnormal |
| | | | | | | | | | | | NCS | CS |
| Day 2 | | | | | | | | | | | | |
| n | | X | | | X | | | X | | | X | |
| Normal | xx | | | | | | | | | | | |
| | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x | (xx.x) | xx (xx.x) | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal | xx | | | | | | | | | | | |
| NCS | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x | (xx.x) | xx (xx.x) | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal | xx | | | | | | | | | | | |
| CS | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x | (xx (xx.x) | xx (xx.x) | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day 15 | | | | | | | | | | | | |
| n | | X | | | X | | | X | | | x | |
| Normal | xx | | | | | | | | | | | |
| | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x | ) xx (xx.x) | xx (xx.x) | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal | xx | | | | | | | | | | | |
| NCS | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x | (xx.x) | xx (xx.x) | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal | XX | | | | | | | | | | | |
| CS | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x | (xx.x) | xx (xx.x) | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

(N)CS = (Not) Clinically Significant.

Baseline is the last non-missing value prior to first dose of study treatment.

Percentages are based on n, the number of subjects with both a baseline and post-baseline result at the study day. Reference: Listing 16.2.8.4

date time

Table 14.3.4.6.2 Summary of QTcF Interval (msec) by Study Day and Result Category (Safety Population)

| Study Day<br>Result Category | GLS-1027<br>120 mg<br>(N=XX) | GLS-1027<br>360 mg<br>(N=XX) | Placebo<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| Baseline | | | | |
| n | x | X | X | x |
| <=450 msec (males) or <=470 msec (females) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >450 msec (males) or >470 msec (females) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day 2 | | | | |
| n | X | X | X | X |
| <=450 msec (males) or <=470 msec (females) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >450 msec (males) or >470 msec (females) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Change from baseline <=60 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Change from baseline >60 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day 15 | | | | |
| n | X | X | X | X |
| <=450 msec (males) or <=470 msec (females) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >450 msec (males) or >470 msec (females) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Change from baseline <=60 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Change from baseline >60 msec | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Baseline is the last non-missing value prior to first dose of study treatment.

Percentages are based on n, the number of subjects with a baseline and post-baseline (for Week 4) result at the study day.

Reference: Listing 16.2.8.4

time date

**APPENDIX D: FIGURE LAYOUTS** 

Protocol: GLS27-005

Figure 14.2.2.1

Line Plot of Mean (+/- SD) PEEP Results During Intubation by Study Day (ITT Population)

Figure 14.2.2.2 Line Plot of Mean (+/- SD) PEEP Results During Intubation by Study Day (PP Population)

Figure 14.3.4.1

Line Plots of Mean (+/-SD) Vital Sign Results by Test and Study Day (Safety Population)

## Figure 14.3.4.2

Line Plots of Mean (+/-SD) 12-Lead ECG Results by Test and Study Day (Safety Population)

APPENDIX E: LISTING LAYOUTS

Listing 16.2.1 Subject Disposition

Treatment: GLS-1027 120 mg

| Subject | Informed | Randomizati | onITT | mITT | Safety | PP | First Dose | Study | Study Completion |
|---|---|---|---|---|---|---|---|---|---|
| ID | Consent<br>Date | Date | Population<br>[1] | Population<br>[2] | Population<br>[3] | Population<br>[4] | Date/Time | Completion<br>Status | or<br>Discontinuation<br>Date<br>(Study Day) |
| xxxx | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | Yes/No | yyyy-mm-dd<br>hh:mm | xxxxxxxxx | yyyy-mm-dd (xx) |
| xxxxx | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | Yes/No | yyyy-mm-dd<br>hh:mm | xxxxxxxxx | yyyy-mm-dd (xx) |
| xxxxx | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | Yes/No | yyyy-mm-dd<br>hh:mm | xxxxxxxxx | yyyy-mm-dd (xx) |
| xxxxx | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | Yes/No | yyyy-mm-dd<br>hh:mm | xxxxxxxxx | yyyy-mm-dd (xx) |
| xxxx | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | Yes/No | yyyy-mm-dd<br>hh:mm | xxxxxxxxx | yyyy-mm-dd (xx) |
| xxxx | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | Yes/No | yyyy-mm-dd<br>hh:mm | xxxxxxxxx | yyyy-mm-dd (xx) |
| xxxx | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | Yes/No | yyyy-mm-dd<br>hh:mm | xxxxxxxxx | yyyy-mm-dd (xx) |
| xxxxx | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | Yes/No | yyyy-mm-dd<br>hh:mm | xxxxxxxxx | yyyy-mm-dd (xx) |

<sup>[1]</sup> The Intent-to-treat (ITT) Population includes all randomized to treatment allocation.

Programming Note: Repeat for each treatment group.

<sup>[2]</sup> The modified intention to treatment (mITT) population includes all participants who are randomized to a treatment allocation, and who have received at least one dose of study drug.

<sup>[3]</sup> The Safety Population includes all subjects who received at least one dose of study drug.

<sup>[4]</sup> The PP Population includes all safety subjects who complete the trial by meeting the endpoint or being discharged within 14 days without meeting the endpoint.

Protocol: GLS27-005

Listing 16.2.2 Protocol Deviations

Treatment: GLS-1027 120 mg

| Deviation Date<br>(Study Day) | Deviation Category | Description |
|---|---|---|
| yyyy-mm-dd (xx) | Major/Minor | XXXXXX |
| yyyy-mm-dd (xx) | Major/Minor | xxxxxx |
| yyyy-mm-dd (xx) | Major/Minor | xxxxxx |
| yyyy-mm-dd (xx) | Major/Minor | xxxxxx |
| yyyy-mm-dd (xx) | Major/Minor | xxxxxx |
| yyyy-mm-dd (xx) | Major/Minor | xxxxxx |
| yyyy-mm-dd (xx) | Major/Minor | xxxxxx |
| yyyy-mm-dd (xx) | Major/Minor | xxxxxx |
| | yyyy-mm-dd (xx) | yyyy-mm-dd (xx) yyyy-mm-dd (xx) Major/Minor |

Programming Note: Repeat for each treatment group.

Listing 16.2.3 Inclusion/Exclusion Criteria

Treatment: GLS-1027 120 mg

| Subject ID | All eligibility criteria met | Criterion not met | Criterion Description |
|---|---|---|---|
| xxxxx | Yes/No | Inclusion xx/Exclusion xx | xxxxxxx |
| XXXXX | Yes/No | Inclusion xx/Exclusion xx | xxxxxxx |
| xxxxx | Yes/No | Inclusion xx/Exclusion xx | xxxxxxx |
| XXXXX | Yes/No | Inclusion xx/Exclusion xx | xxxxxxx |
| xxxxx | Yes/No | Inclusion xx/Exclusion xx | xxxxxxx |
| xxxxx | Yes/No | Inclusion xx/Exclusion xx | xxxxxxx |
| xxxxx | Yes/No | Inclusion xx/Exclusion xx | xxxxxxx |
| XXXXX | Yes/No | Inclusion xx/Exclusion xx | XXXXXXX |

Programming Note: Repeat for each treatment group. If more than one criterion IDs are selected for a subject, list each one on a separate line.

Listing 16.2.4.1
Demographic and Baseline Characteristics

Treatment: GLS-1027 120 mg

| Subject ID | Age<br>(years) | Gender at Birth/<br>Current Gender | Taking Approved Form of Birth Control | Race | Ethnicity | Height<br>(cm) | Weight<br>(kg) | BMI<br>(kg/m^2) |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | XX | Male/Female | Yes | xxxxxxxxxxx | xxxxxxxxxxx | xx.x | xx.x | xx.x |
| xxxxx | XX | Male/Female | No: Reason | xxxxxxxxxxx | XXXXXXXXXXX | xx.x | xx.x | xx.x |
| xxxxx | xx | Male/Female | N/A | xxxxxxxxxxx | xxxxxxxxxxx | xx.x | xx.x | xx.x |
| xxxxx | xx | Male/Female | Yes/No | xxxxxxxxxxx | xxxxxxxxxxx | xx.x | xx.x | xx.x |
| xxxxx | xx | Male/Female | Yes/No | xxxxxxxxxx | xxxxxxxxxxx | xx.x | xx.x | xx.x |

Baseline is the last non-missing value prior to first dose of study treatment.

date time

Programming Note: Repeat for each treatment group.


GeneOne Life Science Inc. Protocol: GLS27-005

Listing 16.2.4.2 Medical History

Treatment: GLS-1027 120 mg

| Subject ID | Any medical history | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date | Ongoing | Stop Date |
|---|---|---|---|---|---|
| xxxxx | Yes/No | xxxxxxxxx/<br>xxxxxxxxx/ | yyyy-mm-dd | Yes/No | yyyy-mm-dd |
| | | xxxxxxxxx<br>xxxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxx | yyyy-mm-dd | Yes/No | yyyy-mm-dd |
| xxxxx | Yes/No | xxxxxxxxx/<br>xxxxxxxxx/ | yyyy-mm-dd | Yes/No | yyyy-mm-dd |
| | | xxxxxxxxx<br>xxxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxx | yyyy-mm-dd | Yes/No | yyyy-mm-dd |
| xxxxx | Yes/No | xxxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxxx | yyyy-mm-dd | Yes/No | yyyy-mm-dd |
| | | xxxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxxx | yyyy-mm-dd | Yes/No | yyyy-mm-dd |

MedDRA = Medical Dictionary for Regulatory Activities.
Medical history terms are coded using MedDRA version 23.0.

Programming Note: Repeat for each treatment group.
Listing 16.2.4.3
Prior and Concomitant Medications

Treatment: GLS-1027 120 mg

| Subject ID | ATC Class/<br>Preferred Name/<br>Verbatim Term | Start Date<br>(Study Day) | End Date<br>(Study Day) | Dose | Units | Route | Frequency | Indication |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxxx | yyyy-mm-dd (xx) | yyyy-mm-dd (xx) | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx |
| | xxxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxx | yyyy-mm-dd (xx) | yyyy-mm-dd (xx) | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx |
| xxxxx | xxxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxxx* | yyyy-mm-dd (xx) | yyyy-mm-dd (xx) | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | xxxxxxxxx | xxxxxxxxx |
| | xxxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxx* | yyyy-mm-dd (xx) | yyyy-mm-dd (xx) | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx |
| ••• | | | | | | | | |

Medications are coded using WHODrug Global (March 2020).

Prior medications are denoted by \*. Prior corticosteroids are denoted by +.

A prior medication is defined as a medication that started and stopped prior to first dose of study treatment. A concomitant medication is any medication that is ongoing or started on or after the date of first dose.

date time

GeneOne Life Science Inc.


Protocol: GLS27-005

Listing 16.2.5.1
Treatment Exposure

Treatment: GLS-1027 120 mg

| Subject ID | Date/time of first dose | Date/time of last dose | Duration of Exposure<br>(days) [1] | Number of Days<br>with At Least<br>One Dose Taken | Total Doses Taken | Total Doses Missed |
|---|---|---|---|---|---|---|
| xxxxx | yyyy-mm-dd hh:mm | yyyy-mm-dd hh:mm | XX | XX | xx | xx |
| xxxxx | yyyy-mm-dd hh:mm | yyyy-mm-dd hh:mm | xx | xx | XX | xx |
| xxxxx | yyyy-mm-dd hh:mm | yyyy-mm-dd hh:mm | xx | xx | xx | xx |
| xxxxx | yyyy-mm-dd hh:mm | yyyy-mm-dd hh:mm | xx | xx | XX | xx |
| xxxxx | yyyy-mm-dd hh:mm | yyyy-mm-dd hh:mm | xx | xx | xx | xx |
| xxxxx | yyyy-mm-dd hh:mm | yyyy-mm-dd hh:mm | xx | xx | XX | xx |
| xxxxx | yyyy-mm-dd hh:mm | yyyy-mm-dd hh:mm | xx | xx | xx | xx |
| xxxxx | yyyy-mm-dd hh:mm | yyyy-mm-dd hh:mm | XX | XX | XX | XX |

<sup>[1]</sup> Duration of exposure is defined as the date of last dose minus the date of first dose + 1.

Listing 16.2.5.2 Study Drug Administration

Treatment: GLS-1027 120 mg

| Subject ID | Study Day | Study drug<br>administered | Date/time of administration | Full dose given | If partial dose,<br>amount given | Number of pills administered |
|---|---|---|---|---|---|---|
| «xxxx | xxxxxx | Yes/No: Reason | yyyy-mm-dd hh:mm | Yes/No | XX | xx |
| | xxxxxx | Yes/No: Reason | yyyy-mm-dd hh:mm | Yes/No | XX | xx |
| xxxxx | xxxxxx | Yes/No: Reason | yyyy-mm-dd hh:mm | Yes/No | xx | xx |
| | xxxxxx | Yes/No: Reason | yyyy-mm-dd hh:mm | Yes/No | xx | xx |
| (XXXX | xxxxxx | Yes/No: Reason | yyyy-mm-dd hh:mm | Yes/No | xx | xx |
| | xxxxx | Yes/No: Reason | yyyy-mm-dd hh:mm | Yes/No | XX | XX |
| xxxx | xxxxxx | Yes/No: Reason | yyyy-mm-dd hh:mm | Yes/No | xx | xx |
| | xxxxxx | Yes/No: Reason | yyyy-mm-dd hh:mm | Yes/No | xx | xx |

time

GeneOne Life Science Inc.

Protocol: GLS27-005

## Listing 16.2.5.3 Pharmacokinetic Assessment

Treatment: GLS-1027 120 mg

| Pre-Treatment<br>1 Hour Post-Dose<br>2 Hours Post-Dose | yyyy-mm-dd hh:mm<br>NOT DONE<br>yyyy-mm-dd hh:mm | xx.x |
|---|---|---|
| | | XX.X |
| 4 Hours Post-Dose<br>8 Hours Post-Dose | yyyy-mm-dd hh:mm<br>yyyy-mm-dd hh:mm | xx.x<br>xx.x |
| Pre-Treatment<br>1 Hour Post-Dose | yyyy-mm-dd hh:mm<br>NOT DONE | xx.x |
| 2 Hours Post-Dose | yyyy-mm-dd hh:mm | xx.x |
| 4 Hours Post-Dose | yyyy-mm-dd hh:mm | xx.x |
| 8 Hours Post-Dose | yyyy-mm-dd hh:mm | XX.X |
| | Pre-Treatment 1 Hour Post-Dose 2 Hours Post-Dose 4 Hours Post-Dose | Pre-Treatment yyyy-mm-dd hh:mm 1 Hour Post-Dose NOT DONE 2 Hours Post-Dose yyyy-mm-dd hh:mm 4 Hours Post-Dose yyyy-mm-dd hh:mm |

Listing 16.2.5.4 Blood Draw

Treatment: GLS-1027 120 mg

| Subject<br>ID | Study<br>Day | Blood for Trough Drug<br>Measurement Collected/<br>Volume Collected | Date/Time of Trough Drug<br>Measurement Collection | Blood for Serum<br>Collected/<br>Volume Collected | Date/Time of Serum<br>Collection | Blood for PBMCs<br>Collected/<br>Volume Collected | Date/Time of PBMCs<br>Collection |
|---|---|---|---|---|---|---|---|
| xxxxx | Day 1 | N/A | | Yes/No/xx | yyyy-mm-dd hh:mm | Yes/No/xx | yyyy-mm-dd hh:mm |
| | Day 2 | Yes/No/xx | yyyy-mm-dd hh:mm | N/A | | N/A | N/A |
| | Day 3 | Yes/No/xx | yyyy-mm-dd hh:mm | N/A | | N/A | N/A |
| | Day 4 | Yes/No/xx | yyyy-mm-dd hh:mm | Yes/No/xx | yyyy-mm-dd hh:mm | Yes/No/xx | yyyy-mm-dd hh:mm |
| | Day 9 | Yes/No/xx | yyyy-mm-dd hh:mm | Yes/No/xx | yyyy-mm-dd hh:mm | Yes/No/xx | yyyy-mm-dd hh:mm |
| | Day 16 | Yes/No/xx | yyyy-mm-dd hh:mm | Yes/No/xx | yyyy-mm-dd hh:mm | Yes/No/xx | yyyy-mm-dd hh:mm |
| | Day 23 | Yes/No/xx | yyyy-mm-dd hh:mm | Yes/No/xx | yyyy-mm-dd hh:mm | Yes/No/xx | yyyy-mm-dd hh:mm |
| | Day 28 | Yes/No/xx | yyyy-mm-dd hh:mm | Yes/No/xx | yyyy-mm-dd hh:mm | Yes/No/xx | yyyy-mm-dd hh:mm |

Protocol: GLS27-005

## Listing 16.2.6.1 WHO Clinical Classification

Treatment: GLS-1027 120 mg

| yyyy-mm-dd<br>yyyy-mm-dd<br>yyyy-mm-dd | x<br>x |
|---|---|
| yyyy-mm-dd<br>yyyy-mm-dd | x<br>x |
| yyyy-mm-dd<br>yyyy-mm-dd | x |
| yyyy-mm-dd | |
| yyyy-mm-dd | |
| yyyy-mm-dd | X |
| vvvv-mm-dd | x |
| yyyy-mm-dd | X |
| | yyyy-mm-dd<br>yyyy-mm-dd<br>\xxxx\xxxxx.sas date time |

Listing 16.2.6.2 Mechanical Ventilation

Treatment: GLS-1027 120 mg

| Subject ID | Study Day | Mechanical Ventilation Used | Date of Mechanical<br>Ventilation | Maximal Daily<br>Level of PEEP<br>(cm) | Maximal Daily<br>Level of Delivered<br>FiO <sub>2</sub><br>(%) |
|---|---|---|---|---|---|
| | David | Va a (Na | | | |
| XXXXXX | Day 1 | Yes/No | yyyy-mm-dd<br> | xxx.x | xxx.x |
| | Day 2 | Yes/No | yyyy-mm-dd | xxx.x | xxx.x |
| | ••• | | | | |
| xxxxxx | Day 1 | Yes/No | yyyy-mm-dd | xxx.x | xxx.x |
| | Day 2 | Yes/No | yyyy-mm-dd | xxx.x | xxx.x |
| | ••• | | | | |
| xxxxx | Day 1 | Yes/No | yyyy-mm-dd | xxx.x | xxx.x |
| | Day 2 | Yes/No | yyyy-mm-dd | xxx.x | XXX.X |
| | ••• | | | | |

Listing 16.2.6.3 Nasal Oxygen  $(O_2)$  Administration

Treatment: GLS-1027 120 mg

| Subject ID | Study Day | Nasal 0 <sub>2</sub> Prescribed | Date of Nasal $0_2$ Administration | $O_2$ Flow Rate (L/min) |
|---|---|---|---|---|
| | | | | · |
| XXXXX | Day 1 | Yes/No | yyyy-mm-dd | xxx.xx |
| | Day 2 | Yes/No | yyyy-mm-dd | xxx.xx |
| | ••• | | | |
| xxxxx | Day 1 | Yes/No | yyyy-mm-dd | xxx.xx |
| | Day 2 | Yes/No | yyyy-mm-dd | xxx.xx |
| | ••• | | | |
| xxxxxx | Day 1 | Yes/No | yyyy-mm-dd | xxx.xx |
| | Day 2 | Yes/No | yyyy-mm-dd | xxx.xx |
| | • • • | | | |

# Listing 16.2.6.4 CPAP Use, ECMO Prescription, ICU Admission

Treatment: GLS-1027 120 mg

| Subject ID | Study Day | CPAP Prescribed | Date of CPAP U | seMaximal Daily Level of End Expiratory Pressure Delivered by CPAP (cm) | Was ECMO<br>prescribed? | Date of ECMO prescription | Was patient<br>admitted to I | Date of ICU<br>CU?Admission |
|---|---|---|---|---|---|---|---|---|
| xxxxx | Day 1 | Yes/No | yyyy-mm-dd | xxx.xx | Yes/No | yyyy-mm-dd | Yes/No | yyyy-mm-dd |
| | Day 2 | Yes/No | yyyy-mm-dd | xxx.xx | Yes/No | yyyy-mm-dd | Yes/No | yyyy-mm-dd |
| xxxxx | Day 1 | Yes/No | yyyy-mm-dd | xxx.xx | Yes/No | yyyy-mm-dd | Yes/No | yyyy-mm-dd |
| | Day 2 | Yes/No | yyyy-mm-dd | xxx.xx | Yes/No | yyyy-mm-dd | Yes/No | yyyy-mm-dd |
| xxxxx | Day 1 | Yes/No | yyyy-mm-dd | xxx.xx | Yes/No | yyyy-mm-dd | Yes/No | yyyy-mm-dd |
| | Day 2 | Yes/No | yyyy-mm-dd | xxx.xx | Yes/No | yyyy-mm-dd | Yes/No | yyyy-mm-dd |

Listing 16.2.6.5
SARS-COV-2 IgM Antibody Titer and Response

Treatment: GLS-1027 120 mg

| Subject ID | Study Day | Date of Assessment | Titer |
|---|---|---|---|
| xxxxxx | Day 1 | yyyy-mm-dd | xxx |
| | Day 7 | yyyy-mm-dd | xxx |
| xxxxxx | Day 1 | yyyy-mm-dd | xxx |
| | Day 7 | yyyy-mm-dd | xxx |
| xxxxxx | Day 1 | yyyy-mm-dd | xxx |
| | Day 7 | yyyy-mm-dd | xxx |
| Source: \\xx\xxx\xxx\x | xxx/xxxxx/xxxxxxxxxxx/xxxx/xxx | x.sas date time | |

Protocol: GLS27-005

Listing 16.2.7.1 Adverse Events

Treatment: GLS-1027 120 mg

| Subject ID | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date<br>(Study Day) | End Date<br>(Study Day) | Severity | Relationship | Action Taken | Serious | Outcome | Study<br>Discontinuation | Treatment<br>Required |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxxxxxxxxxxx/<br>xxxxxxxxxxxxxx/<br>xxxxxxxx | yyyy-mm-dd<br>(xx) | yyyy-mm-dd<br>(xx) | Grade x | xxxxxxxx | xxxxxxxxx | Yes/No | xxxxxxxxx | Yes/No | Yes/No |
| xxxxx | xxxxxxxxxxxxx/ xxxxxxxxxxxxxxxxxxxxxxx | yyyy-mm-dd<br>(xx) | yyyy-mm-dd<br>(xx) | Grade x | xxxxxxxxx | xxxxxxxxx | Yes/No | xxxxxxxxx | Yes/No | Yes/No |
| xxxxx | xxxxxxxxxxxxx/<br>xxxxxxxxxxxxxx/<br>xxxxxxxx | yyyy-mm-dd<br>(xx) | yyyy-mm-dd<br>(xx) | Grade x | xxxxxxxxx | xxxxxxxxx | Yes/No | xxxxxxxxx | Yes/No | Yes/No |

date time

Programming Note: Repeat for each treatment group. Sort by Treatment, Subject ID, AE start date and end date.

Repeat Layout of Listing 16.2.7.1 for:

Listing 16.2.7.3 Adverse Events Leading to Study Discontinuation

Protocol: GLS27-005

## Listing 16.2.7.2 Serious Adverse Events

Treatment: GLS-1027 120 mg

| Subject ID | System Organ Class/<br>Preferred Term/<br>Verbatim Term | | End Date<br>(Study Day) | Severity | Relationship | Action Taken | SAE Criteria | Outcome | Study<br>Discontinuation | Treatment<br>Required |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxxxxxxxxxxx/ xxxxxxxxxxxxxxxxxxxxxxx | yyyy-mm-dd<br>(xx) | yyyy-mm-dd<br>(xx) | Grade x | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxx | Yes/No | Yes/No |
| xxxxx | xxxxxxxxxxxxx/ xxxxxxxxxxxxxxxxxxxxxxx | yyyy-mm-dd<br>(xx) | yyyy-mm-dd<br>(xx) | Grade x | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | Yes/No | Yes/No |
| xxxxx | xxxxxxxxxxxxx/ xxxxxxxxxxxxxxxxxxxxxxx | yyyy-mm-dd<br>(xx) | yyyy-mm-dd<br>(xx) | Grade x | xxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | Yes/No | Yes/No |
| xxxxxx | xxxxxxxxxxxxx/<br>xxxxxxxxxxxxx/<br>xxxxxxxxx | yyyy-mm-dd<br>(xx) | yyyy-mm-dd<br>(xx) | Grade x | xxxxxxxx | xxxxxxxx | xxxxxxxx | xxxxxxxxx | Yes/No | Yes/No |

SAE = Serious Adverse Event

Programming Note: Repeat for each treatment group. Sort by Treatment, Subject ID, AE start date and end date.


GeneOne Life Science Inc. Protocol: GLS27-005

Listing 16.2.7.4 Deaths

Treatment: GLS-1027 120 mg

| Subject ID | Death Date<br>(Study Day) | If Death is Due to Adverse Event, AE # |
|---|---|---|
| xxxxxx | yyyy-mm-dd (xx) | xx |
| xxxxxx | yyyy-mm-dd (xx) | xx |
| xxxxxx | yyyy-mm-dd (xx) | xx |
| xxxxxx | yyyy-mm-dd (xx) | xx |

date

time

Programming Note: Repeat for each treatment group. Sort by Treatment, Subject ID.

GeneOne Life Science Inc.


Protocol: GLS27-005

Listing 16.2.8.1 Hematology

Treatment: GLS-1027 120 mg

| Subject ID | Study Day | Date<br>(Study Day) | Lab Test | Result |
|------------|-------------|---------------------|-----------|--------|
| xxxxxx | Day 0 | yyyy-mm-dd (xx) | xxxxxxxxx | xx.x |
| | | | xxxxxxxxx | xx.x |
| | | | xxxxxxxxx | xx.x |
| | | | xxxxxxxxx | xx.x |
| | | | xxxxxxxxx | xx.x |
| | | | xxxxxxxxx | xx.x |
| | | | xxxxxxxxx | xx.x |
| | | | xxxxxxxxx | xx.x |
| | Study Day 4 | yyyy-mm-dd (xx) | xxxxxxxxx | xx.x |
| | | , , | xxxxxxxxx | xx.x |

Baseline is the last non-missing value prior to first dose of study treatment.

Programming Note: Repeat for each treatment group.

Repeat for Listing 16.2.8.2 Chemistry

GeneOne Life Science Inc.


Protocol: GLS27-005

Listing 16.2.8.3

Vital Signs

Treatment: GLS-1027 120 mg

| Subject | ID Study D | ay Date/Time of Test | Min/Max Systolic BP<br>(mmHg) | Min/Max Diastolic BP<br>(mmHG) | Min/Max Heart Rate<br>(beats/min) | Min/Max<br>Respiratory Rate<br>(breaths/min) | Min/Max Temperature<br>(∘C) |
|---|---|---|---|---|---|---|---|
| xxxxxx | Day 1 | yyyy-mm-dd hh:mm | xx.x | xx.x | xx.x | xx.x | xx.x |
| | Day 2 | yyyy-mm-dd hh:mm | xx.x | xx.x | xx.x | xx.x | xx.x |
| | Day 3 | yyyy-mm-dd hh:mm | xx.x | xx.x | xx.x | xx.x | xx.x |
| | Day 4 | yyyy-mm-dd hh:mm | xx.x | xx.x | xx.x | xx.x | xx.x |
| | Day 5 | yyyy-mm-dd hh:mm | xx.x | xx.x | xx.x | xx.x | xx.x |
| | Day 6 | yyyy-mm-dd hh:mm | xx.x | xx.x | xx.x | xx.x | xx.x |
| | ••• | | | | | | |

Baseline is defined as the last non-missing value prior to the first dose of study treatment. SBP=Systolic Blood Pressure, DBP=Diastolic Blood Pressure.

## Listing 16.2.8.4 12-Lead Electrocardiogram

Treatment: GLS-1027 120 mg

| Subject ID | Study Day | ECG Date/Time | Parameter | Result | Overall Interpretation | Abnormal CS Findings |
|---|---|---|---|---|---|---|
| xxxxx | Hospital Admission | vvvv-mm-dd hh:mm | xxxxxxxxxx | xx.x | Normal/Abnormal NCS/Abnormal CS | xxxxxxxxxxxxxxxx |
| 00000 | Hospital Hamission | <i>yyyy</i> αα | XXXXXXXXXXXX | xx.x | Normal, Normal mai res, Normal mai es | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, |
| | | | XXXXXXXXXXX | XX.X | | |
| | | | XXXXXXXXXXX | XX.X | | |
| | | | XXXXXXXXXXX | xx.x | | |
| | | | xxxxxxxxxxx | xx.x | | |
| | | | xxxxxxxxxxx | xx.x | | |
| | | | xxxxxxxxxx | xx.x | | |
| | Day 2 | yyyy-mm-dd hh:mm | xxxxxxxxxx | xx.x | Normal/Abnormal NCS/Abnormal CS | xxxxxxxxxxxxxxx |
| | • | | xxxxxxxxxx | xx.x | | |
| | | | xxxxxxxxxx | xx.x | | |
| | | | xxxxxxxxxx | xx.x | | |
| | | | XXXXXXXXXXX | xx.x | | |
| | | | XXXXXXXXXXX | xx.x | | |
| | | | XXXXXXXXXXX | XX.X | | |
| | | | XXXXXXXXXXX | xx.x | | |
| | ••• | | | | | |

N(CS)=(Not) Clinically Significant

date time

Protocol: GLS27-005

# Listing 16.2.8.5 Physical Examination

Treatment: GLS-1027 120 mg

| xxxxxx Day 1 Yes/No | yyyy-mm-dd | Yes/No |
|---------------------|------------|--------|
| xxxxxx Day 1 Yes/No | yyyy-mm-dd | Yes/No |
| xxxxxx Day 1 Yes/No | yyyy-mm-dd | Yes/No |
| xxxxxx Day 1 Yes/No | yyyy-mm-dd | Yes/No |

GeneOne Life Science Inc.


Protocol: GLS27-005

Listing 16.2.8.6 Urine Pregnancy Test

Treatment: GLS-1027 120 mg

| Subject ID | Study Day | Test Completed | Date/Time of Test | Result |
|---|---|---|---|---|
| XXXXXX | Day 1 | Yes/No | yyyy-mm-dd | Negative/Positive |
| XXXXXX | Day 1 | Yes/No | yyyy-mm-dd | Negative/Positive |
| XXXXXX | Day 1 | Yes/No | yyyy-mm-dd | Negative/Positive |
| xxxxxx | Day 1 | Yes/No | yyyy-mm-dd | Negative/Positive |
| Source: \\xx\xxx | \xxx\xxx\xxx\x | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | as date time | |

GeneOne Life Science Inc.


Protocol: GLS27-005

Listing 16.2.8.7 Chest X-Ray Score

Treatment: GLS-1027 120 mg

| Study Day | Chest X-Ray Performed | Date of Chest X-Ray | CXR Score |
|---|---|---|---|
| Hospital Admission | Yes/No | yyyy-mm-dd | xxx.xx |
| xxxxx | Yes/No | yyyy-mm-dd | xxx.xx |
| Hospital Admission | Yes/No | yyyy-mm-dd | xxx.xx |
| xxxxx | Yes/No | yyyy-mm-dd | xxx.xx |
| Hospital Admission | Yes/No | yyyy-mm-dd | xxx.xx |
| xxxxx | Yes/No | yyyy-mm-dd | XXX.XX |
| | Hospital Admission xxxxx Hospital Admission xxxxx Hospital Admission | Hospital Admission Yes/No xxxxx Yes/No Hospital Admission Yes/No xxxxx Yes/No Hospital Admission Yes/No | Hospital Admission Yes/No yyyy-mm-dd yxxxxx Yes/No yyyy-mm-dd yyyy-mm-dd yxxxxx Yes/No yyyy-mm-dd yxxxxx Yes/No yyyy-mm-dd yxxxxx Yes/No yyyy-mm-dd yyyyy-mm-dd yyyyy-mm-dd |

## DocuSign<sup>®</sup>

#### **Certificate Of Completion**

Envelope Id: 809EB1C2727A4834A85933CC3530ED1B

Subject: Please DocuSign: GeneOne\_GLS27-005\_SAP\_v1.0\_Catalyst\_03Dec2021.pdf

Source Envelope:

Document Pages: 91 Certificate Pages: 5

AutoNav: Enabled

**Envelopeld Stamping: Disabled** 

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed

Envelope Originator: Ahmed Tariq

5826 Fayetville Rd

Suite 202

Durham, NC 27713

ahmed.tariq@catalystcr.com IP Address: 74.71.122.151

Sent: 12/3/2021 3:21:57 PM

Viewed: 12/3/2021 3:22:31 PM

Signed: 12/3/2021 3:23:17 PM

#### **Record Tracking**

Status: Original

12/3/2021 3:17:54 PM

Holder: Ahmed Tariq

ahmed.tariq@catalystcr.com

Location: DocuSign

**Timestamp** 

#### **Signer Events**

Ahmed Tariq

ahmed.tariq@catalystcr.com

Catalyst Clinical Research - Part 11

Security Level: Email, Account Authentication

(Required)

#### Signature

Signatures: 2

Initials: 0

Ahmed Taria

Signature Adoption: Pre-selected Style

Signature ID:

8A9AFFC7-511B-4804-9134-C7E9728C3D84

Using IP Address: 74.71.122.151

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I am the author of this document

#### **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

Susan E. Spruill

sspruill@appstatsconsulting.com

Security Level: Email, Account Authentication

(Required)

Susan E. Spruill

Sent: 12/3/2021 3:21:57 PM

Viewed: 12/5/2021 8:53:06 AM Signed: 12/5/2021 8:54:12 AM

Signature Adoption: Pre-selected Style

Signature ID:

6B44CB45-B795-4FD5-B700-ED25E98AB084

Using IP Address: 99.197.222.18

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 12/5/2021 8:53:06 AM

ID: e8e1e6ba-5d8e-4116-b669-e9d992005840

| In Person Signer Events | Signature | Timestamp |
|------------------------------|-----------|-----------|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |

| Carbon Copy Events | Status | Timestamp |
|---|---|---|
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 12/3/2021 3:21:57 PM |
| Certified Delivered | Security Checked | 12/5/2021 8:53:06 AM |
| Signing Complete | Security Checked | 12/5/2021 8:54:12 AM |
| Completed | Security Checked | 12/5/2021 8:54:12 AM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disc | osure | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Catalyst Clinical Research - Part 11 (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

## Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

## Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

### **How to contact Catalyst Clinical Research - Part 11:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: shawnegerton@catalystcr.com

### To advise Catalyst Clinical Research - Part 11 of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at shawnegerton@catalystcr.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

## To request paper copies from Catalyst Clinical Research - Part 11

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to shawnegerton@catalystcr.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

## To withdraw your consent with Catalyst Clinical Research - Part 11

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to shawnegerton@catalystcr.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

## Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

## Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Catalyst Clinical Research Part 11 as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by Catalyst Clinical Research Part 11 during the course of your relationship with Catalyst Clinical Research Part 11.